# NCT03078075

# STATISTICAL ANALYSIS PLAN for

Title: NIDA CTN-0068 Accelerated Development of Additive Pharmacotherapy Treatment (ADAPT-2) for Methamphetamine Use Disorder

Version 3.0

Date: September 13, 2019



# Statistical Analysis Plan for NIDA CTN-0068 Protocol

# Accelerated Development of Additive Pharmacotherapy Treatment (ADAPT-2) for Methamphetamine Use Disorder

Lead Investigator: Madhukar Trivedi, MD

Version 3.0 September 13, 2019

Prepared by:
NIDA CTN Data and Statistics Center

## **TABLE OF CONTENTS**

| 1.0 | SUMMARY OF STUDY DESIGN AND PROCESS | 1 |
|-------|----------------------------------------------------|----|
| 1.1 | Study Objective | 1 |
| 1.2 | Study Design and Procedures | 1 |
| 1.2.1 | Study Design | 1 |
| 1.2.2 | Study Procedures | 1 |
| 1.2.3 | Randomization | 2 |
| 1.3 | Inclusion and Exclusion Criteria | 2 |
| 1.3.1 | Inclusion Criteria | 2 |
| 1.3.2 | 2 Exclusion Criteria | 3 |
| 2.0 | GENERAL DEFINITIONS AND PROCEDURES | 4 |
| 2.1 | Pre-screened Population | 4 |
| 2.2 | Screened Population | 4 |
| 2.3 | Randomized Population | 4 |
| 2.4 | Intent-to-Treat Population | 4 |
| 2.5 | Per Protocol Population | 4 |
| 2.6 | Safety Population | 4 |
| 2.7 | Study Day Definition | 4 |
| 2.8 | First Dose Date | 5 |
| 2.9 | Last Dose Date | 5 |
| 2.10 | Treatment Period | 5 |
| 2.11 | Follow-up Period | 5 |
| 2.12 | Safety Window | 5 |
| 2.13 | Treatment Emergence | 5 |
| 2.14 | Summary Table Conventions | 5 |
| 2.15 | Data and Statistics Center Responsibilities | 5 |
| 3.0 | ENROLLMENT, PARTICIPANT DISPOSITION, AND FOLLOW-UP | 6 |
| 4.0 | ANALYSIS OF PARTICIPANT CHARACTERISTICS | 6 |
| 5.0 | CONCOMITANT MEDICATIONS | 6 |
| 6.0 | STUDY MEDICATION ADHERENCE | 7 |
| 6.1 | Early Medication Terminations | 7 |
| 6.2 | Treatment Exposure | 7 |
| 6.3 | Video Confirmed Oral Medication Dosing | 7 |
| 6.4 | Oral Medication Blood Levels | 8 |
| 7.0 | ANALYSIS OF EFFICACY OUTCOME MEASURES | 8 |
| 7.1 | Definition of Primary Outcome Measure | 8 |
| 7.2 | Analysis of Primary Outcome Measure | |
| 7.3 | Supportive Analyses of Primary Outcome Measure | |
| 7.4 | Secondary Outcome Measures | |
| 7.5 | Secondary Outcome Analyses | 11 |

| 8.0 | OTHER STATISTICAL CONSIDERATIONS | 13 |
|---|---|---|
| 8.1 | Handling Missing Data | 13 |
| 8.2 | Significance Testing | 13 |
| 8.3 | Sample Size and Power Calculations | 13 |
| 8.4 | Interim Analyses | 16 |
| 8.4. | Sample Size Re-Estimation | 16 |
| | 8.4.1.1 Sample Size Re-Estimation Results | 17 |
| 8.4.2 | Interim Monitoring of Primary Efficacy Endpoint | 18 |
| 8.4.3 | Safety Interim Analyses | 19 |
| 8.4.4 | Conditional Power and Futility | 20 |
| 8.4.5 | Results of Interim Monitoring for Efficacy and Safety | 20 |
| 8.5 | Software to be Used for Analyses | |
| 9.0 | ANALYSIS OF SAFETY OUTCOME MEASURES | |
| 9.1 | Adverse Events | 20 |
| 9.2 | Serious Adverse Events | |
| 9.3 | Injection Site Abnormalities | |
| 9.4 | Laboratory Values | |
| 9.5 | Electrocardiogram | |
| 9.6 | Suicide Risk | 23 |
| 9.7 | Pregnancy | 23 |
| 9.8 | Deaths | |
| 10.0 | DATA QUALITY | 23 |
| 10.1 | Data Audits | 23 |
| 10.2 | | |
| 11.0 | UPDATES TO THE STATISTICAL ANALYSIS PLAN | 23 |
| 12.0 | REFERENCES | |
| 13.0 | LIST OF PROPOSED TABLES, FIGURES, AND LISTINGS | |
| 14.0 | APPENDICES | 28 |
| 14.1 | Table Shells | 28 |
| | TABLES | |
| Table ' | 1: Secondary Outcomes by Type of Outcome for SPCD Analysis | 12 |
| Table 2 | 2: Primary Outcome Analysis Boundary and Cumulative Alpha Spent | 13 |
| | 3: Sample Size Calculation | |
| Table 4 | 4: Sample Size Re-Estimation Results | 18 |
| Table : | 5: Simulated Probability of Rejecting the Null Hypothesis at $\alpha$ = 0.025, 1-tailed | 19 |
| Table ( | 6: Boundary to Stop Early for Efficacy and Cumulative Alpha Spent at Interim Anal | - |
| Table | 7: Normal Ranges by Site | 22 |
| Table ' | 1: Summary of Pre-screens by Site | 28 |

| Table 2: Summary of Screen Failures by Site | .29 |
|---|---|
| Table 3: Summary of Pre-screens, Screening, and Randomization by Site | . 30 |
| Table 4: Randomizations by Site, Stage and Treatment Arm | .31 |
| Table 5: Proposed and Actual Randomizations by Site | . 35 |
| Table 6: Summary of Disposition by Site | .36 |
| Table 7: Summary of Disposition by Treatment Arm in Stage 1 | .37 |
| Table 8: Summary of Disposition by Treatment Arm in Stage 2 | .38 |
| Table 9: Summary of Disposition by Treatment Arm in Follow-up Period | .39 |
| Table 10: Summary of Attendance at Treatment Period Visits by Treatment Arm in Stage 1. | .41 |
| Table 11: Summary of Attendance at Treatment Period Visits by Treatment Arm in Stage 2. | .42 |
| Table 12: Summary of Attendance at Follow-up Visits by Treatment Arm | .42 |
| Table 13: Summary of Missed Visits by Treatment Arm in Stage 1 | .43 |
| Table 14: Summary of Missed Visits by Treatment Arm in Stage 2 | .44 |
| Table 15: Summary of Missed Visits by Treatment Arm in Follow-up Period | .45 |
| Table 16: Summary of Baseline Characteristics by Site | . 46 |
| Table 17: Summary of Baseline Characteristics by Stage and Treatment Arm | . 50 |
| Table 18: Summary of Concomitant Medications by Treatment Arm <sup>1</sup> | .54 |
| Table 19: Summary of Early Medication Terminations by Site | . 57 |
| Table 20: Summary of Early Medication Terminations by Treatment Arm in Stage 1 | . 59 |
| Table 21: Summary of Early Medication Terminations by Treatment Arm in Stage 2 | .60 |
| Table 22: Summary of Treatment Exposure by Site | .61 |
| Table 23: Summary of Treatment Exposure by Site, Stage and Treatment Arm | .62 |
| Table 24: Summary of Injections by Site | . 64 |
| Table 25: Summary of Injections by Stage and Treatment Arm | . 64 |
| Table 26: Summary of Oral Medication Blood Levels by Stage AMC Participants | .65 |
| Table 27: Summary of Primary Outcome Availability by Stage and Treatment Arm ITT Population | .65 |
| Table 28: Summary of Primary Outcome Analysis by Stage and Treatment Arm ITT Populat | ion |
| | .66 |
| Table 29: Summary of Primary Outcome Sensitivity Analyses by Stage and Treatment Arm ITT Population | .68 |
| Table 30: Summary of Primary Outcome Availability by Stage and Site ITT Population | .69 |
| Table 31: Summary of Primary Outcome by Site, Stage, and Treatment Arm ITT Population | .70 |
| Table 32: Summary of Primary Outcome by Sex, Stage, and Treatment Arm ITT Population. | .70 |
| Table 33: Summary of Primary Outcome by Race, Stage, and Treatment Arm ITT Population | า71 |
| Table 34: Summary of Primary Outcome by Ethnicity, Stage, and Treatment Arm ITT Population | .71 |
| Table 35: Summary of Primary Outcome by Age, Stage, and Treatment Arm ITT Population | .72 |
| Table 36: Primary Outcome Covariate Adjusted Analysis Results <sup>1</sup> ITT Population | .72 |
| Table 37: Summary of UDS Availability <sup>1</sup> by Stage and Treatment Arm Randomized Populati | |
| Table 38: Summary of Methamphetamine Negative UDS Results by Treatment Arm in Stage Randomized Population | |

| Randomized Population75 |
|---|
| Table 40: Summary of Methamphetamine Negative UDS Results by Treatment Arm in Follow-<br>up Period Randomized Population |
| Table 41: Summary of Primary Outcome Sensitivity Analyses by Stage and Treatment Arm Randomized Population |
| Table 42: Summary of Primary Outcome by Stage and Treatment Arm Per Protocol Populations79 |
| Table 43: Summary of Treatment Emergent Adverse Events by Treatment Arm in Stage 180 |
| Table 44: Summary of Treatment Emergent Adverse Events by Treatment Arm in Stage 281 |
| Table 45: Summary of Treatment Emergent MedDRA Coded Adverse Events by Treatment Arm in Stage 182 |
| Table 46: Summary of Treatment Emergent MedDRA Coded Adverse Events by Treatment Arm in Stage 285 |
| Table 47: Summary of Treatment Emergent Serious Adverse Events by Treatment Arm in Stage 197 |
| Table 48: Summary of Treatment Emergent Serious Adverse Events by Treatment Arm in Stage 298 |
| Table 49: Summary of Treatment Emergent MedDRA Coded Serious Adverse Events by Treatment Arm in Stage 199 |
| Table 50: Summary of Treatment Emergent MedDRA Coded Serious Adverse Events by Treatment Arm in Stage 2 |
| Table 51: Summary of Injection Site Abnormalities by Treatment Arm in Stage 1104 |
| Table 52: Summary of Injection Site Abnormalities by Treatment Arm in Stage 2105 |
| Table 53: Summary of Elevated QTc Intervals by Treatment Arm116 |
| Table 54: Summary of Suicide Risk by Treatment Arm in Stage 1120 |
| Table 55: Summary of Suicide Risk by Treatment Arm in Stage 2120 |
| Table 56: Summary of Suicide Risk by Treatment Arm in Follow-up Period120 |
| Table 57: Summary of Data Audits133 |
| Table 58: Summary of Protocol Deviations134 |
| FIGURES |
| Figure 1: SPCD: Defining the Outcome8 |
| Figure 2: Completed Stage 1 and Fraction of Target Enrollment for Proposed Sample Size Re-<br>Estimation Based on Months from Start of Enrollment17 |
| Figure 1: Expected versus Actual Randomizations Overall32 |
| Figure 2: Expected versus Actual Randomizations by Site |
| Figure 2: Expected versus Actual Randomizations by Site (cont.)34 |
| Figure 3: CONSORT Flow Diagram40 |
| Figure 4: Methamphetamine Negative UDS Results by Stage and Treatment Arm ITT Population67 |
| Figure 5: Methamphetamine Negative UDS Results by Stage and Treatment Arm Randomized |
| Population |

# **LISTINGS**

| Listing 1: Treatment Emergent Adverse Events by Treatment Arm | 88 |
|---|---|
| Listing 2: Non-Treatment Emergent Adverse Events in Randomized Participants by<br>Arm | |
| Listing 3: Non-Treatment Emergent Adverse Events in Screen Failure Participants | |
| Listing 4: Serious Adverse Events by Treatment Arm | 101 |
| Listing 5: Injection Site Abnormalities by Treatment Arm | 106 |
| Listing 6: Elevated LFTs by Treatment Arm | 110 |
| Listing 7: Decreased Platelets by Treatment Arm | 114 |
| Listing 8: AV Block ECG Abnormalities by Treatment Arm | 118 |
| Listing 9: Suicide Risk by Treatment Arm | 121 |
| Listing 10: Pregnancies by Treatment Arm | 125 |
| Listing 11: Deaths by Treatment Arm | 129 |
| Listing 12: Listing of Protocol Deviations | 135 |

#### LIST OF ABBREVIATIONS

AE Adverse Event

ALT Alanine Aminotransferase
AST Aspartate Aminotransferase
AMC Active Medication Combination
ATC Anatomical Therapeutic Chemical
CCTN Center for Clinical Trials Network
CHRT Concise Health Risk Tracking

DSC Data and Statistics Center

DSM-5 Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition

DSMB Data and Safety Monitoring Board

ECG Electrocardiogram

EOM End of Medication form

FSR Final Study Report

IN2 Injection Administration 2 form

ITT Intent-to-Treat

LFT Liver Function Test

NIDA National Institute on Drug Abuse

NNT Number Needed to Treat

ODL Oral Study Medication Dosing Log form

PHQ-9 Patient Health Questionnaire-9

PLB Placebo

QOL Quality of Life

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SOC System Organ Class

SPCD Sequential Parallel Comparison Design

STC Study Completion form

TEA Treatment Effectiveness Assessment

TES Treatment Effectiveness Score

TLFB TimeLine Followback
UDS Urine Drug Screen

VAS Visual Analog Craving Scale WHO World Health Organization

XR-NTX Extended-Release Naltrexone (as Vivitrol®)

#### 1.0 SUMMARY OF STUDY DESIGN AND PROCESS

#### 1.1 Study Objective

The primary objective of this study is to evaluate the efficacy of extended-release naltrexone plus bupropion as a combination pharmacotherapy for methamphetamine use disorder. Secondary objectives include assessing the safety of naltrexone plus bupropion and determining the efficacy of the combination pharmacotherapy on other substance use outcomes, on depression symptom scores, and on quality of life ratings.

#### 1.2 Study Design and Procedures

#### 1.2.1 Study Design

This is a double-blind, placebo-controlled, adaptive randomized clinical trial in which 400 individuals with moderate or severe methamphetamine use disorder will be randomly assigned to either 1) active medication combination (AMC) arm in which injections of extended-release naltrexone (XR-NTX; as Vivitrol®) plus once daily oral extended-release bupropion tablets or the 2) matching Placebo (PLB) arm in which injections of placebo and once daily oral placebo tablets will be provided during a 12 week medication phase.

This protocol will utilize a two-stage sequential parallel comparison design (SPCD), originally proposed by Fava et al. (2003), and later revised by Chen et al. (2011). Participants will be randomized to Placebo:AMC in the ratio of **0.74:0.26** in Stage 1 of the study and only Stage 1 placebo non-responders will be re-randomized at the beginning of Stage 2 in a 1:1 ratio. The 12-week medication phase is divided into two stages of approximately equal treatment duration.

The original designed sample size for this study was 370. After the pre-specified sample size reestimation, the Center for Clinical Trials Network (CCTN) approved the increase of the sample size to 400 participants (See Section 8.4.1.1).

#### 1.2.2 Study Procedures

Participants randomized to the AMC arm will receive injections of extended-release naltrexone (Vivitrol®) plus 450 mg of once-daily oral extended-release bupropion tablets while participants randomized to the Placebo arm will receive placebo injections plus once-daily oral placebo tablets. Injectable study medications will be administered every three weeks (Weeks 1, 4, 7, and 10). Take-home oral study medication will be dispensed once weekly for daily dosing. Once weekly medical management sessions with the study medical clinician will be provided. Medication adherence procedures will include smartphone app-confirmation of daily oral study medication dosing using AiCure. Participants will be asked to attend clinic twice weekly for observed oral study medication dosing, collection of urine drug screening samples, and self-report assessments. Compensation will be provided for visit attendance and dosing via AiCure.

Screening/baseline assessments include safety and medical measures including a medical and psychiatric history, a physical examination, clinical lab tests (blood chemistry, hematology, and urinalysis), 12-lead electrocardiogram, vital signs, and pregnancy tests (for females). Screening/baseline assessments also include psychological and drug use measures. Methamphetamine use outcome assessments include Urine Drug Screens (UDS), self-reported use via the Timeline Followback (TLFB), and Visual Analog Scale (VAS) craving scores. Other outcome assessments include UDS and TLFB (i.e., alcohol, tobacco, and/or illicit drugs), depression (Patient Health Questionnaire-9), quality of life (QOL), functioning (Treatment Effectiveness Assessment), and clinic attendance. Safety measures include monitoring vital signs, adverse events (AEs), concomitant medications, clinical lab results, and assessments of suicidality. Oral study medication adherence will be assessed by self-report, quantitative blood

levels of bupropion and its primary metabolite, and smartphone device-based dosing confirmation procedures. A blood sample for genetic analysis will be collected from participants who consent to this procedure and the deidentified sample will be sent to a cell and DNA repository.

At the end of the 12-week medication phase, participants will complete a follow-up phase, including an oral medication taper. Post-medication phase follow-up visits will occur during Weeks 13 and 16. Participants may be withdrawn from study medication for safety reasons due to the discretion of medical clinician. The participant will terminate study medication if there is an increase in liver function tests or a decrease in platelet test results. Refer to Protocol Section 7.2.5 for further information.

#### 1.2.3 Randomization

Eligible participants will be randomized in Stage 1 of the medication phase in a *0.74:0.26* fashion following the SPCD, which is approximately 296:104 participants to the Placebo and AMC treatment arms, respectively (total target N = 400), stratifying by site. Participants who have not been withdrawn from study medication by medical staff will remain eligible to participate in Stage 2. Eligible Stage 1 participants assigned to Placebo and who did not meet the specified definition of responder (i.e., Placebo non-responders) and who attend a visit in the re-randomization window will be re-randomized in a 1:1 ratio to either the Placebo or AMC arm in Stage 2, stratifying by site. All other eligible Stage 1 participants, including participants who did not attend a visit during the re-randomization window, Placebo responders, and AMC participants, will remain in the same treatment arm during Stage 2 as was assigned in Stage 1.

The window for re-randomization opens on Week 7 Day 1 and closes on Week 8 Day 2. If a participant does not attend a visit on or between Week 7 Day 1 and Week 8 Day 2, the participant will not be re-randomized in Stage 2 and will continue receiving the treatment assigned in Stage 1. Re-randomization at Stage 2 helps ensure treatment balance in the two treatment groups within the Stage 2 population.

#### 1.3 Inclusion and Exclusion Criteria

#### 1.3.1 Inclusion Criteria

- 1. 18 to 65 years of age.
- 2. Interested in reducing or stopping methamphetamine use.
- 3. Able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study.
- 4. Meet DSM-5 criteria for moderate or severe methamphetamine use disorder (4 or more criteria.)
- 5. Self-report methamphetamine use on 18 or more days in the 30-day period prior to consent on TLFB.
- 6. Provide at least 2 urine samples positive for methamphetamine out of a possible 3 tests to occur within a 10-day period during which clinic visits occur with at least 2 days between visits.
- 7. If female, agree to use acceptable birth control methods and have periodic urine pregnancy testing done during participation in the study unless documentation of hysterectomy provided.
- 8. Meet subjective and objective measures of being opioid-free prior to naltrexone induction per study medical clinician's determination.
- 9. Willing to comply with all study procedures and medication instructions.

10. Agree to use a smartphone app (downloaded for free to own device or on a study provided smartphone device) to take daily videos of medication dosing.

#### 1.3.2 Exclusion Criteria

- 1. Have an acute medical or psychiatric disorder that would, in the judgment of the study medical clinician, make participation difficult or unsafe.
- 2. Have suicidal or homicidal ideation that requires immediate attention.
- 3. Have a history of epilepsy, seizure disorder, or head trauma with neurological sequelae (e.g., loss of consciousness that required hospitalization); current anorexia nervosa or bulimia; or any other conditions that increase seizure risk in the opinion of the study medical clinician.
- 4. Have evidence of second- or third-degree heart block, atrial fibrillation, atrial flutter, prolongation of the QTc, or any other finding on the screening electrocardiogram (ECG) that, in the opinion of the study medical clinician, would preclude safe participation in the study.
- 5. Have Stage 2 hypertension as determined by the study medical clinician (e.g., greater than or equal to 160/100 in 2 out of 3 readings during screening.)
- 6. Have any elevated bilirubin test value per laboratory criteria OR any other liver function test (LFT) value > 5 times the upper limit of normal per laboratory criteria.
- 7. Have a platelet count <  $100 \times 10^3/\mu$ L.
- 8. Have a body habitus that precludes gluteal intramuscular injection of XR-NTX in accordance with the administration equipment (needle) and procedures.
- Have a known allergy or sensitivity to bupropion, naloxone, naltrexone, PLG (polyactide-co-glycolide), carboxymethylcellulose or any other component of the XR-NTX diluents.
- 10. Have been in a prior study of pharmacological or behavioral treatment for methamphetamine use disorder within 6 months of study consent.
- 11. Have taken an investigational drug in another study within 30 days of study consent.
- 12. Have been prescribed and taken naltrexone or bupropion within 30 days of study consent.
- 13. Concurrently enrolled in formal behavioral or pharmacological addiction treatment services.
- 14. Receiving ongoing treatment with tricyclic antidepressants, xanthines (i.e., theophylline and aminophylline), systemic corticosteroids, nelfinavir, efavirenz, chlorpromazine, MAOIs, central nervous system stimulants (e.g., Adderall, Ritalin, etc.), or any medication that, in the judgment of the study medical clinician, could interact adversely with study medications.
- 15. Have a current pattern of alcohol, benzodiazepine, or other sedative hypnotic use which would preclude safe participation in the study as determined by the study medical clinician.
- 16. Require treatment with opioid-containing medications (e.g., opioid analgesics) during the study period.
- 17. Have a surgery planned or scheduled during the study period.

- 18. Are currently in jail, prison or any inpatient overnight facility as required by court of law or have pending legal action or other situation (e.g., unstable living arrangements) that could prevent participation in the study or in any study activities.
- 19. If female, be currently pregnant, breastfeeding, or planning on conception.

#### 2.0 GENERAL DEFINITIONS AND PROCEDURES

#### 2.1 Pre-screened Population

The pre-screened population consists of all participants who provided verbal consent for the pre-screen process.

#### 2.2 Screened Population

The screened population consists of all participants who provided informed consent at the initiation of the screening process.

#### 2.3 Randomized Population

The Randomized population consists of all participants randomized in Stage 1.

#### 2.4 Intent-to-Treat Population

The Intent-to-Treat (ITT) population consists of all randomized participants in Stage 1. For Stage 2, the ITT population includes all participants who were re-randomized.

#### 2.5 Per Protocol Population

The Per Protocol (PP) population is a subgroup of the ITT population. The PP population consists of participants who have not taken bupropion outside of the study medication, have not taken the incorrect treatment assignment, do not terminate study medication early, meet all entry criteria, complete the treatment period as defined in Section 2.10, and meet treatment exposure requirements. Four PP populations will be defined using the following treatment exposure criteria:

- 1. For each stage, participants who have greater than or equal to 75% treatment exposure for oral study medication and receive 2 injections. Each stage will have its own PP population.
- 2. For each stage, participants who have greater than or equal to 50% treatment exposure for oral study medication and receive at least one injection during the stage. Each stage will have its own PP population.
- 3. For each stage, participants who are greater than or equal to 50% compliant to oral study medication using AiCure confirmed dosing.
- 4. Participants randomized to AMC in Stage 1 who have 2 oral medication blood levels collected during Stage 1 which indicate bupropion dosing, as defined in Section 6.4, and participants re-randomized to AMC in Stage 2 who have 2 oral medication blood levels collected which indicate bupropion dosing. Each stage will have its own PP population.

#### 2.6 Safety Population

The safety population includes all participants who completed informed consent during the screening visit.

#### 2.7 Study Day Definition

Study Day 1 is defined as the day of randomization.

#### 2.8 First Dose Date

The first dose date for oral study medication is the first date on the Oral Study Medication Dosing Log (ODL) on which it is indicated that tablets were taken. The first dose for injectable study medication is the first date an injection was administered on the Injection Administration 2 (IN2) form.

#### 2.9 Last Dose Date

The last dose date for oral study medication is the last day on the ODL form on which it is indicated that tablets were taken. The last dose for injectable study medication is the last date an injection was administered on the IN2 form.

#### 2.10 Treatment Period

The treatment period consists of Study Days 1-84, coinciding with the 12-week medication phase.

#### 2.11 Follow-up Period

The follow-up period consists of two study visits during the post-medication phase occurring at Week 13 and Week 16.

#### 2.12 Safety Window

The safety window begins at the first dose date of either oral or injectable study medication, whichever comes first, and ends either 7 days after the last oral medication dose or 28 days after the last injectable medication, whichever comes last.

#### 2.13 Treatment Emergence

Treatment emergent AEs are defined as AEs with a start date during the safety window.

#### 2.14 Summary Table Conventions

All analyses described in this document for the intent-to-treat population will be summarized over all randomized participants by stages (Stage 1 and 2) and treatment arm. Additionally, some analyses for the intent-to-treat population will also be summarized by site. For all summaries of ITT population, participants will be analyzed according to the treatment arm to which they were randomized regardless of the subsequent sequence of events regarding study drug exposure.

Descriptive summaries of the distribution of continuous variables will be presented with percentiles (median, 25<sup>th</sup> and 75<sup>th</sup> percentiles), and with mean, standard deviation, minimum and maximum. Categorical variables will be summarized in terms of frequencies and/or percentages.

Listings presented by treatment arm will include groups for non-re-randomized Placebo and AMC participants, and re-randomized Placebo and AMC participants (Placebo, Placebo/Placebo, Placebo/AMC, AMC).

#### 2.15 Data and Statistics Center Responsibilities

The CTN's DSC will conduct analyses for the Final Study Report, including those related to the primary outcome measure and the supportive analyses listed in Section 7.3, and the analysis for the primary outcome paper, as discussed by and decided upon by the Lead Node, DSC, and Center for Clinical Trials Network (CCTN). The Lead Node will be responsible for the all secondary outcomes and analyses, the AiCure app-confirmed oral medication dosing described in Section 6.3, and the Per Protocol Population definition #3 detailed in Section 2.5 which uses AiCure treatment exposure information.

#### 3.0 ENROLLMENT, PARTICIPANT DISPOSITION, AND FOLLOW-UP

The number of pre-screens and screens completed and the reasons for ineligibility on prescreening and screening will be summarized by site. Note that participants might be screened twice. For participants who were screened twice, they will only be considered for the second screening.

The distribution of treatment assignments by site and stage will be presented. The trajectory of actual randomizations versus the expected number of randomizations according to the first date of randomization and under the assumption that three participants are expected to be randomized per month per site will be graphed by site and overall. Proposed versus actual randomizations will be summarized by site in a tabular fashion.

Participants are defined as study completers if the Week 16 Follow-up Visit is completed as indicated on the Study Completion (STC) form, and are considered as early study terminations if this visit is not completed. Participant disposition will be summarized by site, treatment arm, and stage for the number of participants completing the study, the number of participants early terminating from the study, and the reasons for early study termination. Early study terminations, using the date of last data collection or date of withdrawn consent on the STC form, will be attributed to Stage 1 if the termination occurred prior to the end of Week 6 (Day 42). Study terminations occurring from Day 43 to Day 84 will be considered to occur in Stage 2, and study terminations occurring after Day 84 will be considered to occur during follow-up.

The CONSORT flow diagram will be generated (Moher et al., 2010).

The number and percentage of participants who attend the bi-weekly treatment period study visits during Weeks 1-12 will be presented by treatment arm and stage, and the Week 13 and 16 follow-up visits will be presented by treatment arm. Information on missed visits during the treatment period and the follow-up period will be presented by treatment arm and stage, including the number of missed visits, the number of participants with at least one missed visit, and the reasons for the missed visits. The expected number of visits during the treatment period is calculated based on the general rule that two visits per week are expected per participant for a total of 12 expected visits per stage, and two visits are expected during the follow-up period. The average number of missed visits per participant will be calculated by dividing the number of missed visits by the number of participants. For early study terminations, visits are only considered missed during active study participation if they occur before the study termination date.

#### 4.0 ANALYSIS OF PARTICIPANT CHARACTERISTICS

Baseline demographics and characteristics including sex, age, ethnicity, race, education level, marital status, employment status, and the number of methamphetamine use days in the 30 days prior to informed consent reported on TLFB will be summarized by site, treatment arm, and stage. Because randomization is expected to produce balance at baseline between the two arms of the trial, statistical comparisons of treatment groups with respect to baseline characteristics will be informal. If differences between treatments arms are suspected, statistical testing will be performed.

#### 5.0 CONCOMITANT MEDICATIONS

Concomitant medications taken during the treatment period will be coded using the WHO Drug Dictionary. Summaries by treatment arm will be presented by Anatomical Therapeutic Chemical (ATC) Class level 1 and ATC Class level 2 and will include the number and percentage of participants receiving each drug class during the safety window defined in Section 2.12.

#### 6.0 STUDY MEDICATION ADHERENCE

Exposure to study medication will be assessed by oral medication dosing, including self-report and AiCure app-confirmed dosing, injection administration, and medication blood levels.

#### **6.1** Early Medication Terminations

Participants may terminate early from either oral study medication or injectable study medication, or from both study medications. Participants will be considered early oral medication terminations as of the date of last oral medication dose entered on the End of Medication (EOM) form. For injectable study medication the date of early medication termination is not collected, and participants will be considered to terminate from the medication for the injection number after the last injection administered on the IN2 form. Early injection termination participants receiving no injections or injection #1 only will be considered early injection terminations in Stage 1, and participants last receiving injection #2 or #3 will be considered early injection terminations in Stage 2. Note there is one exception that participants terminating the study or terminating both study medications on or before Day 42 (end of Week 6) who received both injection #1 and #2 will be considered as early injectable study medication terminations in Stage 1. Early oral study medication terminations occurring before the date of re-randomization or Day 43 for participants who are not re-randomized are considered to occur in Stage 1, and early oral study medications occurring on or after the date of re-randomization are assigned to Stage 2.

The number of participants terminating early from each study medications and the reasons for termination will be presented by site and by stage and treatment arm.

#### 6.2 Treatment Exposure

During the treatment period (Days 1-84), 3 tablets per study day are expected and 4 injections should be administered. Oral study medication dosing is recorded on the ODL form and injection administration is recorded on the IN2 form. Treatment exposure is defined as the average of the percentage of expected oral study medication taken and the percentage of expected injections received. Oral medication taken after the end of the treatment period Day 84 will not be considered. Treatment exposure will be summarized by site, and by site, treatment arm and stage. Oral medication expected to be taken before the date of re-randomization or Study Day 43 for non-re-randomized participants is considered Stage 1, and oral medication expected to be taken on or after the date of re-randomization or Study Day 43 for non-re-randomized participants is considered Stage 2. Injections #1 and #2 are allocated to Stage 1 and injections #3 and #4 are in Stage 2.

A summary of the number of injections administered out of the 4 expected injections by site and by treatment arm and stage will be presented. Two injections are expected in each stage.

#### 6.3 Video Confirmed Oral Medication Dosing

Exposure to oral medication will also be calculated using information from the smartphone appbased dosing confirmation procedures developed by AiCure. Video confirmed dosing adherence data is to be interpreted as an objective indicator of the lowest medication adherence rate participants achieve. Video confirmed adherence is defined as the percentage of expected oral study medication taken, with taken medication including dosing confirmed via video, confirmed by the site, and confirmed in the clinic. Oral medication taken after the end of the treatment period Day 84 will not be considered. Video confirmed adherence will be summarized by site and by treatment arm and stage.

#### 6.4 Oral Medication Blood Levels

Exposure to bupropion will be assessed at Weeks 4, 7, 10, and 12 for participants randomized to AMC and Weeks 10 and 12 for participants re-randomized to AMC by examining quantitative blood levels of bupropion and its primary metabolite hydroxybupropion. Bupropion blood levels greater than 0.500 ng/mL (limit of detection) and hydroxybupropion blood levels greater than 1.00 ng/mL (limit of detection) will indicate adherence to oral bupropion dosing. A summary table of AMC participants adherent to bupropion dosing by stage will be provided.

#### 7.0 ANALYSIS OF EFFICACY OUTCOME MEASURES

#### 7.1 Definition of Primary Outcome Measure

The evaluation period is the final two weeks of the medication phase in Stage 1 (Weeks 5-6) for all participants and Stage 2 (Weeks 11-12) for participants that have been re-randomized. The primary efficacy outcome is a measurement of treatment response at a specified threshold (3 of 4 UDS negative for methamphetamine during the two-week period). Thus, a participant will meet responder criterion by providing 3 or 4 methamphetamine-negative UDS tests during the final two weeks of each stage of the treatment period. All other participants without 3 or 4 methamphetamine-negative UDS will be considered non-responders.

It is hypothesized that the AMC arm will be associated with a greater number of responders, relative to the Placebo arm. The treatment groups will be compared as to the proportion of responders in Stage 1 and Stage 2. The treatment effect will be defined as a weighted combination of the response rates in the two stages. The weight was chosen to optimize the test under the alternative hypothesis as described below. In addition, clinically it is expected that a larger treatment effect will be observed in Stage 2 due to the exclusion of placebo responders from Stage 1. All treatment comparisons will be performed under the Intent-to-Treat (ITT) criteria.

#### 7.2 Analysis of Primary Outcome Measure

Figure 1 shows the design parameters of the SPCD.



Figure 1: SPCD: Defining the Outcome

Let **p1**, **q1** be the response rates for AMC and Placebo in Stage 1; and **p2**, **q2** be the response rates of AMC and Placebo in Stage 2, that is, among Placebo non-responders. Assume that **s** is the rate of continuation into Stage 2 among Placebo non-responders, (i.e., 1-s is the Stage 1 drop-out rate). The primary analysis alternative hypothesis is that the AMC group has higher

response rate than Placebo in the full population (Stage 1) OR in the sub-population of Placebo non-responders (Stage 2). The following null ( $H_0$ ) vs alternate hypothesis ( $H_1$ ) will be tested:

$$H_0$$
:  $p_1 \le q_1$  AND  $p_2 \le q_2$ 

$$H_1: p_1 > q_1 \text{ OR } p_2 > q_2$$

The randomization fraction, a and the weight, w are the parameters of the SPCD that are chosen to maximize the power of the test, based on the alternative hypothesis. Fava (2003) recommends that both a and w be chosen a priori based on the alternative hypothesis of interest. For the alternative hypothesis of this study, it is assumed p1=0.24, q1=0.15 (response rates for AMC and Placebo, respectively, in Stage 1) and p2=0.24, q2=0.10 (response rates for AMC and Placebo, respectively, in Stage 2), and s=0.85 (rate of continuation into Stage 2 of the trial among Placebo non-responders). These assumptions lead to the conclusion that the randomization fraction, a=0.37 and the weight, w=0.43 will maximize the power of the test. The primary outcome analysis will be performed as described in Tamura and Huang (2007) using the Wald type test statistic Z=h/se(h), where

$$h = w(p_{1,obs} - q_{1,obs}) + (1 - w)(p_{2,obs} - q_{2,obs})$$

$$var(h) = \frac{w^{2}p_{1,obs}(1 - p_{1,obs})}{n(1 - 2a)} + \frac{\left(\left(\frac{w^{2}}{4}\right)q_{1,obs}(1 - q_{1,obs}) + \frac{(1 - w)^{2}q_{2,obs}(1 - q_{2,obs})}{s_{obs}(1 - q_{1,obs})}\right)}{na} + \frac{\left(\left(\frac{w^{2}}{4}\right)q_{1,obs}(1 - q_{1,obs}) + \frac{(1 - w)^{2}p_{2,obs}(1 - p_{2,obs})}{s_{obs}(1 - q_{1,obs})}\right)}{na}$$

and 
$$se(h) = \sqrt{var(h)}$$

Note that Schoenfeld corrected the Tamura and Huang formula for the variance.

In the above test statistic both  $\boldsymbol{a}$  and  $\boldsymbol{w}$  are chosen a priori as 0.37 and 0.43; n is the sample size and the quantities  $p_{1,obs}$ ,  $q_{1,obs}$ ,  $s_{obs}$ ,  $p_{2,obs}$  and  $q_{2,obs}$  will be estimated from the data. The null hypothesis will be rejected if Z > boundary (one-sided), where the boundary for interim and final analysis is defined as the O'Brien-Fleming boundary as described in Section 8.4.2. A one-sided p-value for the test of primary outcome will be presented. One-sided lower bound confidence limit for the responder rate will be calculated using h - boundary x se(h). See Section 8.2 for the boundary and cumulative alpha spent to be used at interim analysis and final analysis.

The Number Needed to Treat (NNT) will be calculated as 1/h. UDS availability and results in the evaluation periods will be summarized by treatment arm and stage. A graph of the percentage of negative methamphetamine UDS results during the treatment and follow-up periods will be presented.

#### 7.3 Supportive Analyses of Primary Outcome Measure

The analysis will be repeated with the inclusion of selected covariates, for example, age of onset of methamphetamine use, baseline number of methamphetamine use days self-reported on Timeline Followback (TLFB) in the 30 days prior to informed consent, severity of methamphetamine use (presence or absence of using methamphetamine via injection route of administration on TLFB in the 30 days prior to informed consent; number of DSM-5 criteria met

during screening), tobacco use (number of days using cigarettes or e-cigarette on TLFB during 30 days prior to informed consent), Treatment Effectiveness Assessment score at screening, average of all Visual Analog Craving scale scores collected during screening, and site. A generalized linear mixed effect model will be used to assess the covariate adjusted treatment effects to use in the equation in Section 7.2 to compute h.

Subgroup analysis for sex, race, ethnicity and age will be performed as required by the NIH (NIH, 2016). A generalized linear mixed effect model will be used to assess the subgroup-by-stage-by-treatment interaction. A contrast will be written using the pre-specified weight ( $\mathbf{w}$ =0.43) to test the difference in the primary hypothesis by subgroup.

The primary hypothesis is the difference in the weighted treatment effect in Stage 1 and 2. For example, the difference in the primary hypothesis by sex (Female = F, Male = M) is obtained by a contrast using the weighted treatment effects within males ( $h_M$ ) and females ( $h_F$ ) which are given by the following equations:

$$h_M = \{ w(p_{1,M} - q_{1,M}) + (1 - w)(p_{2,M} - q_{2,M}) \}$$
  
$$h_F = \{ w(p_{1,F} - q_{1,F}) + (1 - w)(p_{2,F} - q_{2,F}) \}$$

The estimates for the responder rate and standard error for males and females will be obtained using an LSMESTIMATE statement and the p-value for the comparison will be obtained using a CONTRAST statement in the SAS code below.

```
proc glimmix data=final method=quad;
  class sex stage trt patid;
  model responder = sex*stage*trt/noint solution;
  random intercept /subject=patid;
  contrast "MvsF" sex*stage*trt -.43 .43 -.57 .57 .43 -.43 .57 -.57;
  lsmestimate sex*stage*trt "Male" -.43 .43 -.57 .57;
  lsmestimate sex*stage*trt "Female" 0 0 0 0 -.43 .43 -.57 .57;
  run;
```

Similarly, the subgroup analysis for site, race, ethnicity, and age will be conducted. If there are more than 2 levels of a subgroup e.g. race (black, white and other) an overall p-value will be reported and appropriate post-hoc testing will be conducted. Summary tables of primary outcome results by site and in the subgroups for sex, race, ethnicity, and age will be provided by treatment arm.

Responder rates in the Randomized Population and the Per Protocol Populations will be presented by treatment arm.

A sensitivity analysis using w=0.5 will be performed for the ITT Population.

#### 7.4 Secondary Outcome Measures

Secondary outcome measures for the impact of the AMC, relative to the Placebo arm, on other substance use outcomes, depression scores, quality of life, overall functioning, clinic attendance, and medication adherence will be evaluated as follows.

- 1. Alternate measures and composites of methamphetamine use including:
  - a) The Treatment Effectiveness Score (TES) (Ling et al., 1997), as measured by UDS results, during the treatment period. The TES is the percentage of the expected urine drug screens that were negative for each drug. Twelve urine drug screens are expected within each stage.

- b) Methamphetamine use, as measured by UDS, during the treatment period. Outcomes include UDS results in the pre-evaluation period (Weeks 1-4 for Stage 1 and Weeks 7-10 in Stage 2), the maximum number of consecutive negative UDS (missing and positive UDS will reset the count to zero), and number of study weeks during the treatment period with two methamphetamine-negative UDS.
- c) Frequency of methamphetamine use, as measured by self-report on TLFB, during the treatment period. The self-reported number of days abstinent from methamphetamine use will be assessed during the evaluation periods during Stage 1 and Stage 2 and over the entire treatment period.
- d) Severity of methamphetamine craving, as measured by Visual Analog Craving Scales (VAS), during the treatment period. VAS scores range from 0 (no craving) to 100 (most intense craving possible). The VAS is completed at screening, once a week during the treatment period, and at the follow-up visits.
- e) Methamphetamine use as measured by UDS and methamphetamine use self-reported on TLFB during the follow-up period. UDS results and the self-reported number of days abstinent from methamphetamine use during the follow-up will be assessed.
- 2. Other substance use, as measured by UDS, during the treatment period. Opioid use will also be assessed using the Opioid 2000 ng tests on the UDS.
- 3. Quantity and frequency of alcohol, quantity and frequency of cigarettes, frequency of ecigarettes, and frequency of other drug use, as measured by self-report on TLFB during the treatment period.
- 4. Depressive symptoms, as measured by the PHQ-9, during the treatment period. The PHQ-9 is collected at screening, once a week during the treatment period, and at the follow-up visits.
- 5. Quality of life (QoL), as measured by the PhenX Core Tier 1 instrument and collected on the Quality of Life (QLP) form, during the treatment period. Ratings of general health, physical health, and mental health during the past 30 days at screening, mid-treatment (Week 6 Visit 2), and end-of-treatment (Week 12 Visit 2) are collected.
- 6. Overall functioning, as measured by the Treatment Effectiveness Assessment (TEA), during the treatment period. The Treatment Effectiveness Assessment (Ling, 2012) is a 4-item self-administered assessment that uses a Likert scale (1-10) to document changes in four life domains: substance use, health, lifestyle, and community and is collected at screening, mid-treatment (Week 6 Visit 2) and end-of-treatment (Week 12 Visit 2).
- 7. Percentage of participants who completed a visit in Week 12.
- 8. Ratings of participant and staff satisfaction with study procedures, including use of the medication adherence app, compensation, and medication.

The Lead Node will provide summary tables by treatment arm and stage for the above secondary outcomes.

#### 7.5 Secondary Outcome Analyses

All secondary analyses described below will be conducted by the Lead Node. The secondary outcomes listed in Section 7.4 are classified in Table 1.

| Table | Table 1: Secondary Outcomes by Type of Outcome for SPCD Analysis | |
|---|---|---|
| Type of Outcome | Frequency of Measurement | Outcomes |
| Binary Cross-<br>Sectional | one<br>measurement per<br>stage | Meth use from UDS (1.b, 1.e) Other substance use from UDS (2) |
| Ordinal | one<br>measurement | Ratings of participant and staff satisfaction (8) |
| Ordinal Cross-<br>Sectional one<br>measurement per<br>stage | | QOL (general health) (5) |
| Count | one<br>measurement per<br>stage | Number of weeks with meth-negative UDS (1.b) Number of consecutive meth-negative UDS (1.b) Number of meth-abstinent TLFB days (1.c, 1.e) Number of alcohol, cigarettes, e-cigarettes, and other substance use TLFB days (3) |
| Continuous | one<br>measurement | Treatment completion (7) |
| Continuous<br>Cross-<br>Sectional | one<br>measurement per<br>stage | TES (1.a) Quantity of alcohol and cigarettes used from TLFB (3) QOL (physical health, mental health) (5) TEA (substance use, health, lifestyle, community) (6) |
| Continuous<br>Repeated<br>Measures | multiple<br>measurements<br>per stage | Severity of meth craving measured by VAS (1.d) PHQ-9 (4) |

Binary cross-sectional outcomes will be analyzed using the same model as for the primary outcome. All repeated measures will be analyzed using the method of Doros et al, 2012. The mixed effects repeated measures models will control for baseline methamphetamine use days self-reported on TLFB and other key demographic and participant variables such as severity of methamphetamine use, tobacco use history, and visual analog craving scale. Nonparametric analyses will be used if the assumptions of the mixed effects analysis cannot be met. Participant and staff satisfaction ratings will be summarized. Analyses of secondary outcomes will be primarily performed on all individuals who are in the ITT population and inducted onto both study medications.

The analysis approach described in Doros et al, 2012 is preferred, however the approach defined in Chen (2011) may also be used, as appropriate (i.e., for continuous outcome ordinary least squares and mixed effects models for repeated measures (MMRM). Logistic regression may also be used for binary outcomes. The same weights as primary outcome will be used to calculate the weighted combination of the estimated treatment effects in the two stages for the secondary analyses.

Secondary analyses of outcomes not specified in Section 7.4 will also be performed. Adherence to oral study medication dosing will be measured by smartphone app-confirmation of daily oral study medication dosing and as recorded on the dosing log (ODL). In addition, per protocol analyses will be conducted using the Per Protocol population definitions in Section 2.5. Because

per protocol analyses may be biased (Sheiner and Rubin, 1995), an unbiased complier-adjusted causal effects analysis (Stuart and Jo, 2015) may also be used to adjust for adherence.

Additionally, methamphetamine and other substance use outcomes may be assessed for responders, non-responders, and other subgroups.

#### 8.0 OTHER STATISTICAL CONSIDERATIONS

#### 8.1 Handling Missing Data

Any participant who drops out before the last week in each evaluation period is, by definition, a non-responder. Therefore, any participant who drops out before Week 6 is a Stage 1 non-responder. In the SPCD design, Stage 1 Placebo non-responders are to be randomized again in Stage 2, but re-randomization is impossible if the participant has dropped out. Thus, Stage 1 dropouts will not contribute to the analysis in Stage 2. In Stage 2, dropouts (i.e., any participant who drops out before Week 12) are again considered to be non-responders by definition, and this causes no further complication in the SPCD computation.

It is unknown *a priori* how many participants will drop out in Stage 1 of the study, thus the 15% attrition rate (**s=0.85**) was chosen as a conservative estimate. Also, as described above, an assumption was made that participants who dropped out early in a given stage will be considered as non-responders in that stage. Therefore, it is important to assess the impact of these missing data assumptions on the primary outcome analysis of the study. A series of sensitivity analyses will be performed to determine how the missing data affects the primary results. Analysis by imputing missing UDS as negative will be conducted, as well as a complete case analysis which includes all participants who have 4 UDS collected in the evaluation period for each stage. Based on the literature review on novel missing data methodology for SPCD, additional secondary analysis may be performed to support the primary outcome analysis.

#### 8.2 Significance Testing

The primary outcome will be evaluated using a one-sided test with a type I error rate of  $\alpha$ =0.025, adjusted based on O'Brien-Fleming boundaries for the interim analysis as described in Section 8.4.2. The boundary and the cumulative alpha spent used for interim and final analysis are noted below in Table 2.

| Table 2: Primary Outcome Analysis Boundary and Cumulative Alpha Spent | | |
|---|---|---|
| Timepoint | Boundary for Declaring<br>Statistical Significance | Alpha Level<br>(Cumulative alpha spent) |
| Interim analysis | 2.9626 | 0.00153 |
| Final analysis | 1.9686 | 0.025 |

The secondary outcomes will use a two-sided test with 5% error rate. There are several secondary outcomes; however, multiple testing will not be adjusted for in the secondary analyses, since these are not part of the study's primary objective. When multiple tests are conducted, the chance of finding a significant difference in one of the tests, when in fact no difference exists, is greater than the stated type I error rate. The investigators are aware of the issues associated with multiple testing and will interpret results with caution.

#### 8.3 Sample Size and Power Calculations

The sample size calculation was conducted as described in Tamura and Huang (2007), with the randomization ratio for Placebo:AMC defined as **2a:(1-2a)**, where **a** is defined as the

randomization fraction. Table 2 shows the impact of various design assumptions on the parameters of the SPCD, the randomization fraction  $\boldsymbol{a}$ , and the weight  $\boldsymbol{w}$  on the sample size. It is important to note that when the rate of discontinuation is 0% ( $\boldsymbol{s}$ =1), the sample size calculation based on Tamura and Huang (2007) gives the same results as Fava et al. (2003) SPCD sample size calculations.

As described in Section 7.2 for the alternate hypothesis, it is assumed *p1=0.24*, *q1=0.15* (response rates for AMC and Placebo, respectively, in Stage 1) and *p2=0.24*, *q2=0.10* (response rates for AMC and Placebo, respectively, in Stage 2), and *s=0.85* (rate of continuation into Stage 2 of the trial among placebo non-responders). Corresponding to these, the randomization fraction *a=0.37* and the weight *w=0.43* would maximize the power of the test (Table 3). A sample size of 370 is chosen for this study and will provide 90% power to detect the weighted difference between the two treatment arms. In Stage 1, the random allocation to Placebo:AMC would be 274:96. Based on the above assumptions, it would be expected that:

- Of the 274 assigned to PLB, 15% (*q1=0.15*) would be Placebo responders while 85% (or 233) would be Placebo non-responders.
- 198 (85% of 233, **s=0.85**) participants would continue to Stage 2.
- In Stage 2, the random allocation to Placebo: AMC would be 99:99.
- During the course of the entire study 195 participants will receive the AMC, with 96 in Stage 1 and 99 in Stage 2.

See Section 8.4.1.1 for an update to the sample size after the sample size re-estimation was conducted.

| Table 3: Sample Size Calculation | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| SPCD Design Assumptions | | | | | | | | |
| Rate o<br>Continuat<br>Response Rates in Stage | | | | | lmį | pact of Ass | sumptions | on |
| AN | ИС | Pl | В | | Parameters Sample Si | | Parameters Sample Siz | |
| Stage 1<br>(p1) | Stage 2<br>(p2) | Stage 1<br>(q1) | Stage 2<br>(q2) | s | а | w | 80%<br>Power | 90%<br>Power |
| 0.29 | 0.29 | 0.15 | 0.15 | 1 | 0.28 | 0.67 | 187 | 250 |
| 0.29 | 0.29 | 0.15 | 0.10 | 1 | 0.35 | 0.46 | 134 | 179 |
| 0.29 | 0.29 | 0.10 | 0.15 | 1 | 0.23 | 8.0 | 105 | 141 |
| 0.29 | 0.29 | 0.10 | 0.10 | 1 | 0.26 | 0.68 | 89 | 119 |
| 0.29 | 0.24 | 0.15 | 0.15 | 1 | 0.24 | 0.78 | 225 | 301 |
| 0.29 | 0.24 | 0.15 | 0.10 | 1 | 0.29 | 0.61 | 174 | 232 |
| 0.29 | 0.24 | 0.10 | 0.10 | 1 | 0.23 | 0.75 | 102 | 136 |
| 0.24 | 0.29 | 0.15 | 0.15 | 1 | 0.36 | 0.45 | 283 | 379 |
| 0.24 | 0.29 | 0.10 | 0.15 | 1 | 0.25 | 0.73 | 160 | 214 |
| 0.24 | 0.29 | 0.10 | 0.10 | 1 | 0.32 | 0.54 | 120 | 161 |
| 0.24 | 0.24 | 0.15 | 0.15 | 1 | 0.28 | 0.67 | 417 | 558 |
| 0.24 | 0.24 | 0.15 | 0.10 | 1 | 0.4 | 0.33 | 246 | 329 |
| 0.24 | 0.24 | 0.10 | 0.15 | 1 | 0.23 | 0.82 | 187 | 250 |
| 0.24 | 0.24 | 0.10 | 0.10 | 1 | 0.27 | 0.67 | 151 | 201 |
| 0.29 | 0.29 | 0.15 | 0.15 | 0.85 | 0.27 | 0.72 | 196 | 262 |
| 0.29 | 0.29 | 0.15 | 0.10 | 0.85 | 0.33 | 0.54 | 147 | 196 |
| 0.29 | 0.29 | 0.10 | 0.15 | 0.85 | 0.22 | 0.82 | 108 | 144 |
| 0.29 | 0.29 | 0.10 | 0.10 | 0.85 | 0.25 | 0.72 | 94 | 125 |
| 0.29 | 0.24 | 0.15 | 0.15 | 0.85 | 0.24 | 0.81 | 230 | 308 |
| 0.29 | 0.24 | 0.15 | 0.10 | 0.85 | 0.28 | 0.66 | 184 | 246 |
| 0.29 | 0.24 | 0.10 | 0.10 | 0.85 | 0.23 | 0.79 | 105 | 140 |
| 0.24 | 0.29 | 0.15 | 0.15 | 0.85 | 0.34 | 0.54 | 313 | 419 |
| 0.24 | 0.29 | 0.10 | 0.15 | 0.85 | 0.25 | 0.77 | 167 | 223 |
| 0.24 | 0.29 | 0.10 | 0.10 | 0.85 | 0.3 | 0.61 | 131 | 175 |
| 0.24 | 0.24 | 0.15 | 0.15 | 0.85 | 0.27 | 0.71 | 439 | 587 |
| 0.24 | 0.24 | 0.15 | 0.10 | 0.85 | 0.37 | 0.43 | 276 | 370 |
| 0.24 | 0.24 | 0.10 | 0.15 | 0.85 | 0.22 | 0.84 | 190 | 254 |
| 0.24 | 0.24 | 0.10 | 0.10 | 0.85 | 0.26 | 0.72 | 158 | 212 |

#### 8.4 Interim Analyses

#### 8.4.1 Sample Size Re-Estimation

Sample size re-estimation analysis will be conducted when approximately half of the participants have been enrolled and have passed the last day available for re-randomization, Week 8 Day 2, and will focus on the nuisance parameter s (rate of continuation into Stage 2 of the trial among Placebo non-responders). This analysis will not reveal the treatment effect observed in the trial at the time of this interim analysis. Fava (2003) suggested that both a and b be a priori chosen to maximize the power of the test based on the alternative hypothesis of interest, and therefore a and b will not be re-estimated. Under the design assumptions of b p1=0.24, q1=0.15, b p2=0.24, q2=0.10, the randomization fraction b and the weight b sample size re-estimation will be performed using the estimated parameter b sample size and whether a sample size increase is warranted.

The timing of the sample size re-estimation is based on a number of factors: recruitment rate. timing of the primary outcome, amount of loss to follow-up, and time to perform the sample size re-estimation. ADAPT-2 will use the graphical tool presented in Figure 2 to assist in assessing the appropriate timing of sample size re-estimation. To illustrate, Figure 2 shows the timing of reestimation when 50% of the participants have completed Stage 1 in the study (0.5 on the red line), assuming enrollment (blue line) in ADAPT-2 of 370 participants over an 18-month period. The time point to perform the sample size re-estimation corresponds to 10.7 months (9 months to enroll 50% participants plus completion of end of re-randomization window at Week 8 Day 2) after enrollment into ADAPT-2 has started, at which point, the study will have enrolled about 58% of the target sample size. If recruitment takes more or less time than expected, modifications can be made to the timing of the sample size re-estimation. The sample size re-estimation will be done only once and done before any interim analysis of the primary outcome is performed. The results of the sample size re-estimation analysis would be presented in a closed session of the DSMB, who will then provide a recommendation to the NIDA CCTN regarding whether the target sample size should be modified. A decision regarding any such modification would be made subsequently by the CCTN, taking into consideration the recommendation of the DSMB.

1.0 1.0 Fraction of Target Enrolled Fraction of Target with Completed Stage 1 0.9 0.9 0.8 0.8 0.7 0.7 Completed Stage 1 of the Study Fraction of Target Enrolled 0.59 Enrollment (+51 Days) at 0.5 Completed Stage 1. N=220 0.6 0.5 Completed Stage 1. N=185 0.5 0.5 0.4 0.4 months to hit 0.5 Completed Stage 0.3 0.3 End of enrollment 0.2 0.2 0.1 0.1 10.7 0.0 0.0 0 12 24

Figure 2: Completed Stage 1 and Fraction of Target Enrollment for Proposed Sample Size Re-Estimation Based on Months from Start of Enrollment

#### 8.4.1.1 Sample Size Re-Estimation Results

The NIDA CTN DSMB reviewed the sample size re-estimation report dated July 23, 2018, prepared by the DSC. In this report, the sample size re-estimation was presented under the design assumptions of p1=0.24, q1=0.15, p2=0.24, q2=0.10, the randomization fraction a=0.37, the weight w=0.43, and using the estimated parameter s=0.75758, keeping the other parameters fixed. The s parameter was estimated using the first 185 participants randomized. Table 4 shows the results of the sample size re-estimation.

Months from Start of Enrollment

| Table 4: Sample Size Re-Estimation Results | | | |
|---|---|---|---|
| Sample Size Calculation s N Power | | | |
| O interest designs | 0.85 | 276 | 80% |
| Original design | 0.85 | 370 | 90% |
| Power with current | 0.75758 | 276 | 76.8% |
| sample size and updated s parameter | 0.75758 | 370 | 87.7% |
| Maintaining original | 0.75758 | 298 | 80% |
| power with increased sample size using updated <b>s</b> parameter | 0.75758 | 399 | 90% |

Based on the above results, the DSMB and NIDA CCTN concurred that although the loss of power compared to the original power calculations was negligible, the dropout rate that will occur in Stage 2 of the study is also unknown and recommended increasing the sample size by 30 additional participants (N = 400) to maintain the targeted 90% power. The CCTN approved the increase the sample size to 400 participants in a letter to the Lead Investigator dated August 13, 2018.

#### 8.4.2 Interim Monitoring of Primary Efficacy Endpoint

Interim monitoring for efficacy will be performed of the primary alternative hypothesis that the AMC, relative to the Placebo, is associated with greater methamphetamine non-use. There will be no interim efficacy monitoring before a sample size re-estimation is performed (or a determination that re-estimation is not needed) because sample size re-estimation could change the target sample size, affecting the alpha spending function used in the interim efficacy monitoring. After sample size re-estimation, interim efficacy monitoring will be performed only once during the recruitment period. Because the Lan-DeMets approach (DeMets and Lan, 1994) requires an independent increments process, care must be taken in defining the population that will be used in the interim analysis. For example, including participants in an interim look who completed 6 weeks of Stage 1 and are Placebo non-responders, but have not yet had the opportunity to contribute Stage 2 responses, violates the independent-increments requirement. To avoid this, the following rule will be obeyed:

• For a look at study time *t* months, include only those participants who were randomized to Stage I no later than *t*-3 months (i.e., have the opportunity to complete the 12 weeks (or 3 months) on study at the time of the analysis). The size of that sample, when divided by the target sample size, becomes the information fraction for the look at calendar time *t*.

Based on the above rule and using designed parameters, the Lan-DeMets alpha-spending approach to interim monitoring for SPCD trials was investigated by simulation. Enrollment was assumed to be constant over an 18-month period. Under the null hypothesis, (p1, p2) are set equal to (q1, q2) = (0.15, 0.10), while under the alternative, (p1, p2) = (0.24, 0.24) a 2-look scenario, in which information fraction = (0.5, 1.0), was simulated.

Table 5 gives the simulated probability of rejecting the null hypothesis at alpha = 0.025, 1-tailed, for each of these scenarios. More specifically, 10,000 time series of SPCD z-values were simulated, each with 2 values (when there are 2 looks) for each scenario. In each scenario, the proportion of time series that ever cross the relevant boundary is presented in Table 6. It shows that after using the O'Brien-Fleming-type boundaries the test size under the null and power under the alternative are as desired.

| Table 5: Simulated Probability of Rejecting the Null Hypothesis at $\alpha$ = 0.025, 1-tailed | | |
|---|---|---|
| | Alternative<br>Hypothesis | |
| O'Brien-Fleming type | 0.0237 | 0.90 |

All interim monitoring will use an O'Brien-Fleming-type boundary with information fraction equal to the proportion of the target sample size with primary outcome, and alpha = 0.025, one-tailed. This approach spends very little alpha at the interim look, therefore the impact of an interim monitoring on the sample size is negligible. Table 6 shows an example of boundary (Z-score) to stop early for efficacy and cumulative alpha spent at interim analysis with 0.5 information fraction.

| Table 6: Boundary to Stop Early for Efficacy and Cumulative Alpha Spent at Interim Analysis | | | |
|---|---|---|---|
| Information Fraction Boundary Alpha Spent Cumulative Alpha Spen | | | |
| 0.5 (Half-way) | 2.9626 | 0.00153 | 0.00153 |
| 1 (End of study) | 1.9686 | 0.02347 | 0.025 |

In addition, the observed parameters and number of participants assigned to each treatment arm in the two stages will be monitored against the designed parameters (*p1=0.24*, *q1=0.15*, *p2=0.24*, *q2=0.10*, *s=0.85*) and expected assignment. The only criterion for early stopping for efficacy will be based on Z-scores and its relation to O'Brien-Fleming-type boundary.

Before recommending early termination, the DSMB should consider:

- Internal consistency of primary and secondary results.
- Internal consistency of primary and secondary results by subgroups defined by baseline characteristics (e.g., number of baseline MA use days on TLFB, severity of MA use, tobacco use history, treatment effectiveness assessment and visual analog craving scale).
- Distribution of baseline prognostic factors among the two groups.
- Consistency of primary and secondary results across clinical sites and among clinical sites enrolling larger numbers of participants.
- Possible impact of missing data from missed participant visits for assessment of the primary and secondary response variables.
- Possible differences in concomitant interventions or medications.

#### 8.4.3 Safety Interim Analyses

Safety interim looks will be performed for the regular DSMB meetings or at unscheduled times per the DSMB's request. These will include analysis of adverse events and narrative report on serious adverse events.

Further, because the primary outcome analysis is a one-sided test to assess whether AMC is more efficacious than Placebo, simultaneous with primary interim efficacy monitoring analysis, a poor efficacy statistic will be calculated to assess whether the AMC, relative to the Placebo, is associated with greater methamphetamine use i.e., whether compared to AMC, the response rate

is greater in Placebo in both stages. This analysis will be conducted after the sample size reestimation. If the poor efficacy of AMC statistic crosses its boundary, defined by the minimum of q1 - p1 and q2 - p2 being greater than 10%, the DSMB will consider whether to stop the trial early because of poor efficacy of AMC relative to Placebo. When reporting results of the trial, the one-sided superiority test will be considered the primary outcome, with the other tail considered as part of the poor efficacy analysis intended for the DSMB to monitor for safety. That is, as in a more usual trial design, the possibility of exit in the safety/poor efficacy tail will not be considered as possibly affecting the type I or type II error of the primary outcome statistical test.

#### 8.4.4 Conditional Power and Futility

Unless otherwise requested, a futility/conditional power calculation will be performed when interim monitoring is performed. If at any DSMB meeting the conditional power falls below 0.3 (when hypothetical future observations are generated under the design alternative (*p1=0.24*, *q1=0.15*, *p2=0.24*, *q2=0.10*) but tested under the null), this will stimulate a discussion among the DSMB members about whether the trial should stop for futility.

#### 8.4.5 Results of Interim Monitoring for Efficacy and Safety

The NIDA CTN DSMB met on October 24, 2018 to review the interim efficacy and safety analyses prepared by the DSC using the first 200 enrollment participants. The DSMB recommended the study should continue until 400 participants complete as determined by the sample size reestimation.

#### 8.5 Software to be Used for Analyses

The O'Brien-Fleming boundaries and the p-value for the primary outcome will be calculated in WinLD (Reboussin 2000). The interim analyses for sample size re-estimation and conditional power will be conducted in R Versions 3.4.2 and 3.5.1. All other analyses performed by the DSC and the Lead Node will use SAS® Version 9.4 software, including the calculation of the Wald type test statistic Z for the primary outcome. The Lead Node may also conduct analyses using R Versions 3.4.2 and 3.5.1.

#### 9.0 ANALYSIS OF SAFETY OUTCOME MEASURES

#### 9.1 Adverse Events

Treatment emergent adverse events (AEs) as defined in Section 2.13 will be summarized by presenting the number of events, number of participants experiencing AEs, and the severity and relatedness of adverse events by treatment arm and stage. Stage 1 events include AEs occurring before the date of re-randomization for re-randomized participants and in Weeks 1-6 for non-re-randomized participants, and Stage 2 AEs include events occurring on or after the date of re-randomization for re-randomized participants and in Weeks 7 or greater for non-re-randomized participants.

All adverse events will be coded using MedDRA® dictionary version 22.0 and higher and the number of participants experiencing each treatment emergent AE and the incidence rate will be provided by treatment arm and stage. Treatment emergent adverse event incidence rates will be summarized by System Organ Class (SOC) and Preferred Term (PT). The incidence rate of an AE is calculated as the number of participants who experience the event at least once during the safety window divided by the number of participants at risk times 100. Incidence rates will be calculated at the preferred term level, at the SOC level, and for participants with at least one treatment emergent adverse event. If a participant experiences multiple episodes of an event, then the event is only counted once. Detailed listings of treatment emergent adverse events and non-treatment emergent events in the safety population by treatment arm will be provided.

Treatment arm differences will be monitored by the DSMB.

#### 9.2 Serious Adverse Events

Treatment emergent Serious Adverse Events (SAEs) will be summarized by presenting the number of events, number of participants experiencing SAEs, and the relatedness and type of SAEs by treatment arm and stage. SAEs will be presented by stage as described in Section 9.1. A summary of treatment emergent MedDRA® coded serious adverse events using incidence rates will be provided by treatment arm and stage. Incidence rates, as defined in Section 9.1, will be calculated at the preferred term level, at the SOC level, and for participants with at least one treatment emergent serious adverse event. A detailed listing of SAEs, including treatment emergent SAEs and non-treatment emergent SAEs, will be provided by treatment arm. Narratives for all serious adverse events will be included in the Final Study Report.

#### 9.3 Injection Site Abnormalities

The injection site is examined by medical personnel at the next study visit following the injection administration. Injections #1 and #2 occur in Stage 1 and injections #3 and #4 occur in Stage 2. Injection site abnormalities will be summarized by presenting the number of abnormalities, number of participants experiencing abnormalities, type of abnormality, and the severity of the abnormality by treatment arm and stage. A detailed listing of injection site abnormalities for injections by treatment arm will be provided.

#### 9.4 Laboratory Values

Laboratory values are collected at Screening, Week 6, and Week 12. Elevated liver function tests (LFTs) consisting of alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin and decreased platelets are monitored by the safety and medical monitors at the CCC. There are multiple site- and sex-based normal ranges amongst the eight sites for the ALT, AST and total Bilirubin parameters. For practicality, the safety team reviewed these parameters and generated a global threshold for each: ALT and AST 250 IU/L, total bilirubin 2.2 mg/dL, and platelets below 75 x  $10^3/\mu$ L. Table 7 provides the normal ranges for all study sites for LFTs and platelets.

Listings of elevated LFTs and decreased platelets will be presented by treatment arm.

| | | | Table 7: N | Iormal Ranges | by Site | | | |
|---|---|---|---|---|---|---|---|---|
| Lab | SC BHS | WS CODA, Inc. | GNY SURC -<br>Columbia | NS Hennepin<br>County | WS SURU -<br>SFDPH | TX UCLA<br>CBAM | TX UT Health<br>CNRA | TX<br>UTSW |
| ALT | female 14-54<br>IU/L<br>male 17-63 IU/L | Female 16-19 yrs 5-<br>32 U/L<br>Female 20+ yrs 6-<br>29 U/L<br>Male 16-19 yrs 8-46<br>U/L<br>Male 20+ yrs 9-46<br>U/L | Female 1-31 IU/L<br>Male 1-40 IU/L | Female up to 33<br>U/L<br>Male up to 41<br>U/L | Female 7-35 U/L<br>Male 10-40 U/L | 8-64 units/L | Female 0-32<br>IU/L<br>Male 0-44 IU/L | 9-46 U/L |
| AST | 15-41 IU/L | Female 7-19 yrs 12-<br>32 U/L<br>Female 20-49 yrs<br>10-30 U/L<br>Female 50+ yrs 10-<br>35 U/L<br>Male 7-19 yrs 12-32<br>U/L<br>Male 20-49 yrs 10-<br>40 U/L<br>Male 50+ yrs 10-35<br>U/L | Female 1-31 IU/L<br>Male 1-37 IU/L | 5-40 U/L | 2-60 yrs 10-41 U/L<br>60-90 yrs 10-48<br>U/L | 13-47 units/L | 0-40 IU/L | 10-40<br>U/L |
| Total<br>Bilirubin | 0.3-1.2 mg/dL | Female 10-19 yrs<br>0.2-1.1 mg/dL<br>Female 20+ yrs 0.2-<br>1.2 mg/dL<br>Male 10-19 yrs 0.2-<br>1.1 mg/dL<br>Male 20+ yrs 0.2-1.2<br>mg/dL | 0.1-1.1 mg/dL | 0.0-1.2 mg/dL | 0-60 years 0.1-1.2<br>mg/dL<br>60-90 yrs 0.1-1.1<br>mg/dL | 0.1-1.2<br>mg/dL | 0.0-1.2 mg/dL | 0.2-1.2<br>mg/dL |
| Platelets | 130-450 x<br>thousand<br>cells/µL | 140-400<br>thousand/µL | 130-400 K/mm <sup>3</sup> | 150-400 x 10 <sup>3</sup><br>µL | 150,000-<br>400,000/mcL | 143-398 x<br>10 <sup>3</sup> /µL | 150-379 x<br>10³/μL | 140-400<br>x10 <sup>3</sup> µL |

#### 9.5 Electrocardiogram

Electrocardiograms (ECG) are conducted at screening and at Week 12. A summary table displaying the count and frequency of participants with elevated QTc intervals greater than and equal to 500 milliseconds and changes from baseline will be presented by treatment arm. Participants experiencing second or third degree AV block at Week 12 will be listed by treatment arm.

#### 9.6 Suicide Risk

The Concise Health Risk Tracking (CHRT) and Patient Health Questionnaire-9 (PHQ-9) surveys are conducted at screening, weekly during the treatment period, and at follow-up visits to assess suicide risk. A summary table of participants endorsing suicidality on either assessment during the treatment period will be presented by treatment arm and stage. A listing of visits where suicidality was endorsed by a participant will be generated.

Endorsement for the CHRT is defined as answering agree or strongly agree to any of the following: (1) I have been having thoughts of killing myself, (2) I have thoughts about how I might kill myself, or (3) I have a plan to kill myself. On the PHQ-9, a participant is considered to have endorsed suicidality if they indicate several days, more than half the days, and nearly every day having thoughts they are better off dead or of hurting themselves.

#### 9.7 Pregnancy

A listing of pregnancies and pregnancy outcomes in randomized participants will be generated. Narratives will also be provided.

#### 9.8 Deaths

A listing of deaths and narratives of deaths will be provided.

#### 10.0 DATA QUALITY

#### 10.1 Data Audits

A summary of data audit results from site interim monitoring visits conducted by CCC monitors will be presented by site.

#### 10.2 Protocol Deviations

Protocol deviations will be summarized by site and will include the number of deviations reported, the number of participants each deviation affects, frequencies for the types of protocol deviations, and information on whether the protocol deviation was deemed minor or major. A detailed listing of protocol deviations by deviation category will be provided.

#### 11.0 UPDATES TO THE STATISTICAL ANALYSIS PLAN

The Statistical Analysis Plan (SAP) Version 0.1 was reviewed by the IRB and DSMB prior to the initiation of the study and contains unblinded information on the study design not included in the protocol. SAP Version 1.0 was updated to include all information necessary for interim analyses to be conducted and was finalized on July 5, 2018. SAP Version 2.0, which included a correction to the formula for standard error for the primary outcome analysis, was finalized on September 6, 2018 before interim analyses were conducted for the October 24, 2018 DSMB meeting. SAP Version 3.0 was finalized prior to data lock to include the remaining information necessary to analyze the study.

SAP Version 0.1 is included in Appendix 14.2 and a detailed Change Log from SAP Version 0.1 to SAP Version 2.0 is located in Appendix 14.3.

#### 12.0 REFERENCES

Chen, Y. F., Yang, Y., Hung, H. M., & Wang, S. J. (2011). Evaluation of performance of some enrichment designs dealing with high placebo response in psychiatric clinical trials. *Contemp Clin Trials*, 32(4), 592-604. doi:10.1016/j.cct.2011.04.006.

DeMets DL, Lan KK. (1994). Interim analysis: the alpha spending function approach. *Stat Med*,13:1341-1356.

Doros, G., Pencina, M., Rybin, D., Meisner, A., Fava, M. (2013). A repeated measures model for analysis of continuous outcomes in sequential parallel comparison design studies, *Statistics in Medicine*, 32:2767-2789.

Fava, M., Evins, A. E., Dorer, D. J., & Schoenfeld, D. A. (2003). The problem of the placebo response in clinical trials for psychiatric disorders: culprits, possible remedies, and a novel study design approach. *Psychother Psychosom*, *72*(3), 115-127. doi:69738.

Ling, W., Shoptaw, S., Wesson, D., Rawson, R. A., Compton, M., & Klett, C. J. (1997). Treatment effectiveness score as an outcome measure in clinical trials. *NIDA Res Monogr*, 175, 208-220.

Moher D, Hopewell S, Schulz KF, Montori V, Gøtzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. (2010). CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. *J Clin Epi*, 63(8): e1-e37.

National Institutes of Health (NIH). (2016). Guidelines for the Review of Inclusion on the Basis of Sex/Gender, Race, Ethnicity, and Age in Clinical Research. https://grants.nih.gov/grants/peer/guidelines\_general/Review\_Human\_subjects\_Inclusion.pdf.

Reboussin DM, DeMets DL, Kim KM, Lan KK. (2000). Computations for group sequential boundaries using the Lan-DeMets spending function method. *Control Clin Trials*, 2000 Jun;21(3):190-207.

Schoenfeld D. Power calculator for a Sequential Parallel Comparison Design (SPCD). http://hedwig.mgh.harvard.edu/biostatistics/node/43

Shiener, L.B., Rubin, D.B. (1995). Intention-to-treat analysis and the goals of clinical trials. *Clinical Pharmacology and Therapeutics*, 57(1):6-15.

Stuart, E.A., Jo, B. (2015). Assessing the sensitivity of methods for estimating principal causal effects, *Statistical Methods in Medical Research*. 24(6) (2015) 657-674.

Tamura, R. N., & Huang, X. (2007). An examination of the efficiency of the sequential parallel design in psychiatric clinical trials. *Clin Trials*, *4*(4), 309-317.

### 13.0 LIST OF PROPOSED TABLES, FIGURES, AND LISTINGS

The listing of tables below contains the tables, figures, and listings which will be provided by the DSC.

| Section | ection Title | |
|---|---|---|
| Enrollment,<br>Participant<br>Disposition, and<br>Follow-up | Summary of Pre-screens by Site | Pre-screened |
| | Summary of Screen Failures by Site | Screened |
| | Summary of Pre-screens, Screening, and Randomization by Site | Pre-screened |
| | Randomizations by Site, Stage and Treatment Arm | ITT |
| | Figure of Expected versus Actual Randomizations Overall | Randomized |
| | Figure of Expected versus Actual Randomizations by Site | Randomized |
| | Proposed and Actual Randomizations by Site | Randomized |
| | Summary of Disposition by Site | Randomized |
| | Summary of Disposition by Treatment Arm in Stage 1 | Randomized |
| | Summary of Disposition by Treatment Arm in Stage 2 | Randomized |
| | Summary of Disposition by Treatment Arm in Follow-up Period | Randomized |
| | CONSORT Flow Diagram | Pre-screened |
| | Summary of Attendance at Treatment Period Visits by Treatment Arm in Stage 1 | Randomized |
| | Summary of Attendance at Treatment Period Visits by Treatment Arm in Stage 2 | Randomized |
| | Summary of Attendance at Follow-up Visits by Treatment Arm | Randomized |
| | Summary of Missed Visits by Treatment Arm in Stage 1 | Randomized |
| | Summary of Missed Visits by Treatment Arm in Stage 2 | Randomized |
| | Summary of Missed Visits by Treatment Arm in Follow-up Period | Randomized |
| Participant | Summary of Baseline Characteristics by Site | Randomized |
| Characteristics at Baseline | Summary of Baseline Characteristics by Stage and Treatment Arm | Randomized |
| Concomitant<br>Medications | Summary of Concomitant Medications by Treatment Arm | Randomized |
| Treatment Exposure | Summary of Early Medication Terminations by Site | Randomized |
| | Summary of Early Medication Terminations by Treatment Arm in Stage 1 | m in Randomized |
| | Summary of Early Medication Terminations by Treatment Arm in Stage 2 | Randomized |
| | Summary of Treatment Exposure by Site | Randomized |

| Section | Title | Population |
|---|---|---|
| | Summary of Treatment Exposure by Site, Stage and Treatment Arm | Randomized |
| | Summary of Injections by Site | Randomized |
| | Summary of Injections by Stage and Treatment Arm | Randomized |
| | Summary of Oral Medication Blood Levels in AMC Participants by Stage | Randomized |
| Primary Outcome | Summary of Primary Outcome Availability by Stage and Treatment Arm | ITT |
| | Summary of Primary Outcome Analysis by Stage and Treatment Arm | ITT |
| | Figure of UDS Results by Stage and Treatment Arm | ITT |
| ı | Summary of Primary Outcome Sensitivity Analyses by Stage and Treatment Arm | ITT |
| | Summary of Primary Outcome Availability by Stage and Site | ITT |
| | Summary of Primary Outcome by Site, Stage, and Treatment Arm | ITT |
| | Summary of Primary Outcome by Sex, Stage, and Treatment Arm | ITT |
| | Summary of Primary Outcome by Race, Stage, and Treatment Arm | ITT |
| | Summary of Primary Outcome by Ethnicity, Stage, and Treatment Arm | ITT |
| | Summary of Primary Outcome by Age, Stage, and Treatment Arm | ITT |
| | Primary Outcome Covariate Adjusted Analysis Results | ITT |
| | Summary of UDS Availability by Stage and Treatment Arm | Randomized |
| | Summary of Methamphetamine Negative UDS Results by Treatment Arm in Stage 1 | Randomized |
| | Summary of Methamphetamine Negative UDS Results by Treatment Arm in Stage 2 | Randomized |
| | Summary of Methamphetamine Negative UDS Results by Treatment Arm in Follow-up Period | Randomized |
| | Summary of Primary Outcome Sensitivity Analyses by Stage and Treatment Arm in the Randomized Population | Randomized |
| | Figure of UDS Results by Stage and Treatment Arm in Randomized Population | Randomized |
| | Summary of Primary Outcome by Stage and Treatment Arm in Per Protocol Populations | Per Protocol |
| Safety Outcomes | Summary of Treatment Emergent Adverse Events by Treatment Arm in Stage 1 | Safety |
| | Summary of Treatment Emergent Adverse Events by Treatment Arm in Stage 2 | Safety |

| Section | Title | Population |
|---|---|---|
| | Summary of Treatment Emergent MedDRA Coded Adverse Events by Treatment Arm in Stage 1 | Safety |
| | Summary of Treatment Emergent MedDRA Coded Adverse Events by Treatment Arm in Stage 2 | Safety |
| | Listing of Treatment Emergent Adverse Events by Treatment Arm | Safety |
| | Listing of Non-Treatment Emergent Adverse Events in Randomized Participants by Treatment Arm | Safety |
| | Listing of Non-Treatment Emergent Adverse Events in Screen Failure Participants | Safety |
| | Summary of Treatment Emergent Serious Adverse Events by Treatment Arm in Stage 1 | Safety |
| | Summary of Treatment Emergent Serious Adverse Events by Treatment Arm in Stage 2 | Safety |
| | Summary of Treatment Emergent MedDRA Coded Serious<br>Adverse Events by Treatment Arm in Stage 1 | Safety |
| | Summary of Treatment Emergent MedDRA Coded Serious Adverse Events by Treatment Arm in Stage 2 | Safety |
| | Listing of Serious Adverse Events by Treatment Arm | Safety |
| | Summary of Injection Site Abnormalities by Treatment Arm in Stage 1 | Safety |
| | Summary of Injection Site Abnormalities by Treatment Arm in Stage 2 | Safety |
| | Listing of Injection Site Abnormalities by Treatment Arm | Safety |
| | Listing of Elevated LFTs by Treatment Arm | Safety |
| | Listing of Decreased Platelets by Treatment Arm | Safety |
| | Summary of Elevated QTc Intervals by Treatment Arm | Safety |
| | Listing of AV Block ECG Abnormalities by Treatment Arm | Safety |
| | Summary of Suicide Risk by Treatment Arm in Stage 1 | Safety |
| | Summary of Suicide Risk by Treatment Arm in Stage 2 | Safety |
| | Summary of Suicide Risk by Treatment Arm in Follow-up Period | Safety |
| | Listing of Suicide Risk by Treatment Arm | Safety |
| | Listing of Pregnancies by Treatment Arm | Safety |
| | Listing of Deaths by Treatment Arm | Safety |
| Data Quality | Summary of Data Audits | N/A |
| Protocol Dovictions | Summary of Protocol Deviations | N/A |
| Protocol Deviations | Listing of Protocol Deviations | |

#### 14.0 APPENDICES

#### 14.1 Table Shells

| Table 1: Summary of Pre-screens by Site | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | SC<br>BHSPC | WS CODA,<br>Inc. | GNY<br>SURC -<br>Columbia | NS<br>Hennepin<br>Healthcare | WS SURU -<br>SFDPH | TX<br>UCLA<br>CBAM | TX UT<br>Health<br>CNRA | TX UTSW | Total |
| Number of pre-screens | N | | | | | | | | |
| Number of ineligible pre-screens | N (%) | | | | | | | | |
| Criteria resulting in ineligibility <sup>1</sup> : | | | | | | | | | |
| Have medical/mental health conditions require monitoring/care/medication | N (%) | | | | | | | | |
| Taking meds for medical/mental health condition | | | | | | | | | |
| Cannot refrain from opioid use | | | | | | | | | |
| Currently enrolled in addiction treatment services | | | | | | | | | |
| Taken naltrexone/bupropion within the last 30 days | | | | | | | | | |
| Not used methamphetamine in the past 30 days | | | | | | | | | |
| Methamphetamine use days in the past 30 days (mean (SD)) | | | | | | | | | |
| Not interested in study or willing to use study meds | | | | | | | | | |
| No current methamphetamine use | | | | | | | | | |
| Not willing to attend 2x week for 12 weeks | | | | | | | | | |
| Age < 18 or Age > 65 | | | | | | | | | |
| No interest in reducing/stopping methamphetamine use | | | | | | | | | |
| Unwilling to use app | | | | | | | | | |
| Currently pregnant or breastfeeding | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Percentages are calculated based on the denominator of the number of ineligibles and may exceed 100% if multiple ineligibility criteria are met for potential participants.
| | SC<br>BHSPC | WS<br>CODA,<br>Inc. | GNY SURC -<br>Columbia | NS Hennepin<br>Healthcare | WS SURU -<br>SFDPH | TX UCLA<br>CBAM | TX UT<br>Health<br>CNRA | TX UTSW | Total |
|---|---|---|---|---|---|---|---|---|---|
| Number consented | N | | | | | | | | |
| Number of screen failures | N (%) | | | | | | | | |
| Failed the following eligibility criteria <sup>1</sup> | | | | | | | | | |
| Meth use on 18+/30 day | N (%) | | | | | | | | |
| Comply with study procedures | | | | | | | | | |
| 2/3 positive meth urine in 10 days | | | | | | | | | |
| Conditions that increase seizure risk | | | | | | | | | |
| Medical/psychiatric disorder | | | | | | | | | |
| ECG finding | | | | | | | | | |
| Stage 2 hypertension | | | | | | | | | |
| Current alcohol/benzo use | | | | | | | | | |
| Opioid-free | | | | | | | | | |
| Elevated bilirubin/LFT 5x ULN | | | | | | | | | |
| Taking contraindicated meds | | | | | | | | | |
| Pregnant/breastfeeding | | | | | | | | | |
| Agrees to use birth control and do urine pregnancy testing | | | | | | | | | |
| DSM-5 meth use disorder | | | | | | | | | |
| Agrees to record videos | | | | | | | | | |
| Platelets< 100 x 10 <sup>3</sup> μL | | | | | | | | | |
| Prescribed and taken study drugs | | | | | | | | | |
| Surgery planned/scheduled | | | | | | | | | |
| Jail | 1 | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Percentages are calculated based on the denominator of the number of ineligibles and may exceed 100% if multiple ineligibility criteria are met for potential participants.

| Ta | able 3: Su | mmary of Pr | e-screens, S | creening | g, and Rai | ndomization | by Site | |
|---|---|---|---|---|---|---|---|---|
| Site | Number<br>of<br>Screens | Percent of<br>Eligible Pre-<br>Screens<br>Screened | Average Number of Days Between Pre-Screen and Scheduled Screening Appointment | Number<br>of<br>Screen<br>Fails | Percent<br>of<br>Screens<br>Who<br>Screen<br>Fail | Number<br>Randomized | Percent of<br>Eligible Pre-<br>Screens<br>Randomized | Percent of<br>Screens<br>Randomized |
| SC BHSPC | N | % | X.X | Ν | % | N | % | % |
| WS CODA, Inc. | | | | | | | | |
| GNY SURC - Columbia | | | | | | | | |
| NS Hennepin Healthcare | | | | | | | | |
| WS SURU - SFDPH | | | | | | | | |
| TX UCLA CBAM | | | | | | | | |
| TX UT Health CNRA | | | | | | | | |
| TX UTSW | | | | | | | | |
| Total | | | | | | | | |

| Table 4: Randomizations | by Site, S | Stage ar | nd Treatm | ent Arm |
|---|---|---|---|---|
| | Stage 1 | | | ge 2<br>domized |
| | Placebo | AMC | Placebo/<br>Placebo | Placebo/<br>AMC |
| SC BHSPC | N (%) | | | |
| WS CODA, Inc. | | | | |
| GNY SURC - Columbia | | | | |
| NS Hennepin Healthcare | | | | |
| WS SURU - SFDPH | | | | |
| TX UCLA CBAM | | | | |
| TX UT Health CNRA | | | | |
| TX UTSW | | | | |
| Total | | | | |



Figure 3: Expected versus Actual Randomizations Overall



Figure 4: Expected versus Actual Randomizations by Site



Figure 5: Expected versus Actual Randomizations by Site (cont.)

| | Table 5: I | Proposed and A | ctual Randomi | zations by Site | | |
|---|---|---|---|---|---|---|
| Site | Proposed<br>Randomization | Date Site Opened for Enrollment | Date of First<br>Randomization | Actual<br>Randomizations | Actual/<br>Proposed<br>(%) | Date of Last<br>Randomization |
| SC BHSPC | N | | | N | % | |
| WS CODA, Inc. | | | | | | |
| GNY SURC - Columbia | | | | | | |
| NS Hennepin Healthcare | | | | | | |
| WS SURU - SFDPH | | | | | | |
| TX UCLA CBAM | | | | | | |
| TX UT Health CNRA | | | | | | |
| TX UTSW | | | | | | |
| Total | | | | | | |

| | | 1410 | 01117 | No | 14/0 | <b>T</b> \/ | TV | | |
|---|---|---|---|---|---|---|---|---|---|
| | SC<br>BHSPC | WS<br>CODA,<br>Inc. | GNY<br>SURC -<br>Columbia | NS<br>Hennepin<br>Healthcare | WS<br>SURU -<br>SFDPH | TX<br>UCLA<br>CBAM | TX UT<br>Health<br>CNRA | TX<br>UTSW | Total |
| Number of participants randomized | Ν | | | | | | | | |
| Number of study completers <sup>1</sup> | N (%) | | | | | | | | |
| Number of early study terminations | N (%) | | | | | | | | |
| Reasons for early study termination | | | | | | | | | |
| Participant failed to return to site and unable to contact | N (%) | | | | | | | | |
| Participant withdrew consent/assent | | | | | | | | | |
| Participant stopped participation due to practical problems | | | | | | | | | |
| Participant moved from area | | | | | | | | | |
| Participant incarcerated | | | | | | | | | |
| Participant terminated due to AE/SAE | | | | | | | | | |
| Participant terminated for other clinical reasons | | | | | | | | | |
| Participant had a significant psychiatric risk | | | | | | | | | |
| Participant deceased | | | | | | | | | |
| Participant terminated due to protocol deviation | | | | | | | | | |
| Participant became pregnant | | | | | | | | | |
| Participant reports intolerable symptoms or side effects | | | | | | | | | |
| Participant reports use of medication that could adversely interact with study medication | | | | | | | | | |
| Clinical deterioration: New onset of psychiatric or medical condition | | | | | | | | | |
| Clinical deterioration: Worsening of pre-existing psychiatric or medical condition | | | | | | | | | |
| Clinical deterioration: Worsening of substance use disorder | | | | | | | | | |
| Clinical deterioration: Overdose | | | | | | | | | |
| Participant terminated for other reason | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Participants who completed the study (Week 16) as reported on the Study Completion (STC) form.

| Table 7: Summary of Disposition by Treatment Arm in Stage 1 | | | |
|---|---|---|---|
| | Placebo | AMC | Total |
| Number of participants randomized | N | | |
| Number of participants who completed Stage 1 <sup>1</sup> | N (%) | | |
| Number of participants re-randomized at the end of Stage 1 | N (%) | | |
| Number of early study terminations in Stage 1 | N (%) | | |
| Reasons for early study termination in Stage 1 | | | |
| Participant failed to return to site and unable to contact | N (%) | | |
| Participant withdrew consent/assent | | | |
| Participant stopped participation due to practical problems | | | |
| Participant moved from area | | | |
| Participant incarcerated | | | |
| Participant terminated due to AE/SAE | | | |
| Participant terminated for other clinical reasons | | | |
| Participant had a significant psychiatric risk | | | |
| Participant deceased | | | |
| Participant terminated due to protocol deviation | | | |
| Participant became pregnant | | | |
| Participant reports intolerable symptoms or side effects | | | |
| Participant reports use of medication that could adversely interact with study medication | | | |
| Clinical deterioration: New onset of psychiatric or medical condition | | | |
| Clinical deterioration: Worsening of pre-existing psychiatric or medical condition | | | |
| Clinical deterioration: Worsening of substance use disorder | | | |
| Clinical deterioration: Overdose | | | |
| Participant terminated for other reason | | | |

<sup>&</sup>lt;sup>1</sup> Participants who did not early terminate from the study in Weeks 1-6.

| | Re-rand | lomized | Not Re-rai | | |
|---|---|---|---|---|---|
| | Placebo/<br>Placebo | Placebo/<br>AMC | Placebo | AMC | Total |
| Number of participants randomized | N | | | | |
| Number of participants in Stage 2 <sup>1</sup> | N | | | | |
| Number of participants that completed Week 12 <sup>2</sup> | N (%) | | | | |
| Number of early study terminations in Weeks 7-12 | N (%) | | | | |
| Reasons for early study termination in Weeks 7-12 | | | | | |
| Participant failed to return to site and unable to contact | N (%) | | | | |
| Participant withdrew consent/assent | | | | | |
| Participant stopped participation due to practical problems | | | | | |
| Participant moved from area | | | | | |
| Participant incarcerated | | | | | |
| Participant terminated due to AE/SAE | | | | | |
| Participant terminated for other clinical reasons | | | | | |
| Participant had a significant psychiatric risk | | | | | |
| Participant deceased | | | | | |
| Participant terminated due to protocol deviation | | | | | |
| Participant became pregnant | | | | | |
| Participant reports intolerable symptoms or side effects | | | | | |
| Participant reports use of medication that could adversely interact with study medication | | | | | |
| Clinical deterioration: New onset of psychiatric or medical condition | | | | | |
| Clinical deterioration: Worsening of pre-existing psychiatric or medical condition | | | | | |
| Clinical deterioration: Worsening of substance use disorder | | | | | |
| Clinical deterioration: Overdose | | | | | |

<sup>&</sup>lt;sup>1</sup> Participants who completed Stage 1 (Weeks 1-6) and were re-randomized or were not re-randomized in Stage 2.

<sup>&</sup>lt;sup>2</sup> Participants who did not early terminate from the study on the STC form in Weeks 7-12.

| Table 9: Summary of Disposition by Treatm | nent Arm i | n Follow-ı | ıp Period | | |
|---|---|---|---|---|---|
| | Re-rand | lomized | Not Re-ran | ndomized | |
| | Placebo/<br>Placebo | Placebo/<br>AMC | Placebo | AMC | Total |
| Number of participants randomized | N | | | | |
| Number of participants who entered the Follow-up Period <sup>1</sup> | | | | | |
| Number of participants who completed the study | | | | | |
| Number of early study terminations in Follow-up Period <sup>2</sup> | N (%) | | | | |
| Reasons for early study termination in Follow-up Period | | | | | |
| Participant failed to return to site and unable to contact | N (%) | | | | |
| Participant withdrew consent/assent | | | | | |
| Participant stopped participation due to practical problems | | | | | |
| Participant moved from area | | | | | |
| Participant incarcerated | | | | | |
| Participant terminated due to AE/SAE | | | | | |
| Participant terminated for other clinical reasons | | | | | |
| Participant had a significant psychiatric risk | | | | | |
| Participant deceased | | | | | |
| Participant terminated due to protocol deviation | | | | | |
| Participant became pregnant | | | | | |
| Participant reports intolerable symptoms or side effects | | | | | |
| Participant reports use of medication that could adversely interact with study medication | | | | | |
| Clinical deterioration: New onset of psychiatric or medical condition | | | | | |
| Clinical deterioration: Worsening of pre-existing psychiatric or medical condition | | | | | |
| Clinical deterioration: Worsening of substance use disorder | | | | | |
| Clinical deterioration: Overdose | | | | | |
| Participant terminated for other reason | | | | | |

<sup>&</sup>lt;sup>1</sup> Participants who completed the treatment period (Week 12).

<sup>&</sup>lt;sup>2</sup> Participants who early terminated from the study in Weeks 13-16



40

| Table 1 | Table 10: Summary of Attendance at Treatment Period Visits by Treatment Arm in Stage 1 | | |
|---|---|---|---|
| Visit | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Visit 0101 | N (%) | | |
| Visit 0102 | | | |
| Visit 0201 | | | |
| Visit 0202 | | | |
| Visit 0301 | | | |
| Visit 0302 | | | |
| Visit 0401 | | | |
| Visit 0402 | | | |
| Visit 0501 | | | |
| Visit 0502 | | | |
| Visit 0601 | | | |
| Visit 0602 | | | |
| Overall | | | |

| | Re-rand | lomized <sup>1</sup> | Not Re-rar | ndomized | |
|---|---|---|---|---|---|
| Visit | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Visit 0701 | N (%) | | | | |
| Visit 0702 | | | | | |
| Visit 0801 | | | | | |
| Visit 0802 | | | | | |
| Visit 0901 | | | | | |
| Visit 0902 | | | | | |
| Visit 1001 | | | | | |
| Visit 1002 | | | | | |
| Visit 1101 | | | | | |
| Visit 1102 | | | | | |
| Visit 1201 | | | | | |
| Visit 1202 | | | | | |
| Overall | | | | | |

<sup>&</sup>lt;sup>1</sup> Participants may be re-randomized at Visit 0701, 0702, or 0801.

| Table 12 | 2: Summary o | of Attendance | e at Follow-u <sub>l</sub> | p Visits by Tr | eatment Arm | |
|---|---|---|---|---|---|---|
| | Re-randomized Not Re-randomized | | Re-randomized | | Re-randomized Not Re-randomized | ndomized |
| Visit | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) | |
| Visit 1301 | N (%) | | | | | |
| Visit 1601 | | | | | | |
| Overall | | | | | | |

| Table 13: Summary of Missed Visits by Treatmer | nt Arm in S | tage 1 | |
|---|---|---|---|
| | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Number of expected visits in Stage 1 <sup>1</sup> | N | | |
| Number of missed visits in Stage 1 due to early study termination | N (%) | | |
| Number of missed visits during active Stage 1 participation | N (%) | | |
| Number of participants with at least one missed visit during active Stage 1 participation | N (%) | | |
| Average number of missed visits in Stage 1 per participant | X.X | | |
| Reason for missed visit | | | |
| Participant failed to return to site and unable to contact | N (%) | | |
| Participant unable to attend visit | | | |
| Participant withdrew consent | | | |
| Other | | | |
| Site closed | | | |
| Participant incarcerated | | | |
| Participant on vacation | | | |
| Participant in hospital, in-patient, or residential treatment | | | |
| Participant illness | | | |
| Participant moved from area | | | |
| Participant deceased | | | |

<sup>&</sup>lt;sup>1</sup> Two visits per week are expected per participant in Weeks 1-6.

| Table 14: Summary of Missed Visits by | Treatmen | t Arm in S | tage 2 | | |
|---|---|---|---|---|---|
| | Re-rand | domized | Not Re-ra | ndomized | |
| | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Number of expected visits in Stage 2¹ | N | | | | |
| Number of missed visits in Stage 2 due to early study termination | N (%) | | | | |
| Number of missed visits during active Stage 2 participation | N (%) | | | | |
| Number of participants with at least one missed visit during active Stage 2 participation | N (%) | | | | |
| Average number of missed visits in Stage 2 per participant | X.X | | | | |
| Reason for missed visit | | | | | |
| Participant failed to return to site and unable to contact | N (%) | | | | |
| Participant unable to attend visit | | | | | |
| Participant withdrew consent | | | | | |
| Other | | | | | |
| Site closed | | | | | |
| Participant incarcerated | | | | | |
| Participant on vacation | | | | | |
| Participant in hospital, in-patient, or residential treatment | | | | | |
| Participant illness | | | | | |
| Participant moved from area | | | | | |
| Participant deceased | | | | | |

<sup>&</sup>lt;sup>1</sup> Two visits per week are expected per participant in Weeks 7-12.

| Table 15: Summary of Missed Visits by Treatm | ent Arm i | n Follow-u | ıp Period | | |
|---|---|---|---|---|---|
| | Re-rand | domized | Not Re-rai | ndomized | |
| | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Number of expected visits in follow-up period¹ | N | | | | |
| Number of missed visits in follow-up period due to early study termination | N (%) | | | | |
| Number of missed visits during active follow-up period participation | N (%) | | | | |
| Number of participants with at least one missed visit during active follow-up period participation | N (%) | | | | |
| Average number of missed visits in follow-up period per participant | X.X | | | | |
| Reason for missed visit | | | | | |
| Participant failed to return to site and unable to contact | N (%) | | | | |
| Participant unable to attend visit | | | | | |
| Participant withdrew consent | | | | | |
| Other | | | | | |
| Site closed | | | | | |
| Participant incarcerated | | | | | |
| Participant on vacation | | | | | |
| Participant in hospital, in-patient, or residential treatment | | | | | |
| Participant illness | | | | | |
| Participant moved from area | | | | | |
| Participant deceased | | | | | |

<sup>&</sup>lt;sup>1</sup> Two visits total are expected per participant in the follow-up period in Weeks 13-16.

| | | | of Baseline | ı | <del>-</del> | | | <u> </u> | |
|---|---|---|---|---|---|---|---|---|---|
| Characteristic | SC<br>BHSPC<br>(N=) | WS<br>CODA,<br>Inc.<br>(N=) | GNY SURC -<br>Columbia<br>(N=) | NS<br>Hennepin<br>Healthcare<br>(N=) | WS SURU -<br>SFDPH<br>(N=) | TX<br>UCLA<br>CBAM<br>(N=) | TX UT<br>Health<br>CNRA<br>(N=) | TX UTSW<br>(N=) | Total<br>(N=) |
| Sex | | | | | | | | | |
| Missing | N (%) | | | | | | | | |
| Male | | | | | | | | | |
| Female | | | | | | | | | |
| Participant chose not to answer | | | | | | | | | |
| Age (Mean (SD)) | XX (X.X) | | | | | | | | |
| Age | | | | | | | | | |
| Missing | N (%) | | | | | | | | |
| < 18 | | | | | | | | | |
| 18 - < 25 | | | | | | | | | |
| 25 - < 35 | | | | | | | | | |
| 35 - < 45 | | | | | | | | | |
| 45 - < 55 | | | | | | | | | |
| 55 - < 65 | | | | | | | | | |
| 65 - < 75 | | | | | | | | | |
| 75+ | | | | | | | | | |
| Ethnicity | | | | | | | | | |
| Missing | | | | | | | | | |
| Not Hispanic or Latino | N (%) | | | | | | | | |
| Hispanic or Latino | | | | | | | | | |
| Participant chose not to answer | | | | | | | | | |

| Т | able 16: S | Summary | of Baseline | Characteris | stics by Site | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Characteristic | SC<br>BHSPC<br>(N=) | WS<br>CODA,<br>Inc.<br>(N=) | GNY SURC -<br>Columbia<br>(N=) | NS<br>Hennepin<br>Healthcare<br>(N=) | WS SURU -<br>SFDPH<br>(N=) | TX<br>UCLA<br>CBAM<br>(N=) | TX UT<br>Health<br>CNRA<br>(N=) | TX UTSW<br>(N=) | Total<br>(N=) |
| Race | | | | | | | | | |
| Missing | N (%) | | | | | | | | |
| American Indian or Alaska Native | | | | | | | | | |
| Asian | | | | | | | | | |
| Black or African American | | | | | | | | | |
| Native Hawaiian or Pacific Islander | | | | | | | | | |
| White | | | | | | | | | |
| Other | | | | | | | | | |
| Multiracial | | | | | | | | | |
| Unknown | | | | | | | | | |
| Participant chose not to answer | | | | | | | | | |
| Education completed | | | | | | | | | |
| Missing | N (%) | | | | | | | | |
| Less than high school diploma | | | | | | | | | |
| High school graduate | | | | | | | | | |
| GED or equivalent | | | | | | | | | |
| Some college, no degree | | | | | | | | | |
| Associate's degree: occupational, technical, or vocational program | | | | | | | | | |
| Associate's degree: academic program | | | | | | | | | |
| Bachelor's degree | | | | | | | | | |
| Master's degree | | | | | | | | | |

| Ta | able 16: S | Summary | of Baseline | Characteris | stics by Site | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Characteristic | SC<br>BHSPC<br>(N=) | WS<br>CODA,<br>Inc.<br>(N=) | GNY SURC -<br>Columbia<br>(N=) | NS<br>Hennepin<br>Healthcare<br>(N=) | WS SURU -<br>SFDPH<br>(N=) | TX<br>UCLA<br>CBAM<br>(N=) | TX UT<br>Health<br>CNRA<br>(N=) | TX UTSW (N=) | Total<br>(N=) |
| Professional school degree | | | | | | | | | |
| Doctoral degree | | | | | | | | | |
| Don't know | | | | | | | | | |
| Refused | | | | | | | | | |
| Marital status | | | | | | | | | |
| Missing | N (%) | | | | | | | | |
| Married | | | | | | | | | |
| Widowed | | | | | | | | | |
| Divorced | | | | | | | | | |
| Separated | | | | | | | | | |
| Never married | | | | | | | | | |
| Living with partner | | | | | | | | | |
| Refused | | | | | | | | | |
| Don't know | | | | | | | | | |
| Employment | | | | | | | | | |
| Missing | N (%) | | | | | | | | |
| Working now | | | | | | | | | |
| Only temporarily laid off, sick leave, or maternity leave | | | | | | | | | |
| Looking for work, unemployed | | | | | | | | | |
| Retired | | | | | | | | | |
| Disabled permanently or temporarily | | | | | | | | | |

| Та | able 16: S | Summary | of Baseline | Characteris | stics by Site | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Characteristic | SC<br>BHSPC<br>(N=) | WS<br>CODA,<br>Inc.<br>(N=) | GNY SURC -<br>Columbia<br>(N=) | NS<br>Hennepin<br>Healthcare<br>(N=) | WS SURU -<br>SFDPH<br>(N=) | TX<br>UCLA<br>CBAM<br>(N=) | TX UT<br>Health<br>CNRA<br>(N=) | TX UTSW (N=) | Total<br>(N=) |
| Keeping house | | | | | | | | | |
| Student | | | | | | | | | |
| Other | | | | | | | | | |
| Number of days of self-reported methamphetamine use in 30 days prior to informed consent | | | | | | | | | |
| N | | | | | | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| Min | | | | | | | | | |
| 25th Percentile | | | | | | | | | |
| Median | | | | | | | | | |
| 75th Percentile | | | | | | | | | |
| Max | | | | | | | | | |

| Table 17: Summary o | of Baseline Characteristi | cs by S | tage and Tr | eatment Arı | m | |
|---|---|---|---|---|---|---|
| | | | Stage 2 | | | |
| | Stag | e 1 | Re-ran | domized | Not Re-ra | ndomized |
| Characteristic | Placebo<br>(N=) | AMC<br>(N=) | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) |
| Sex | | | | | | |
| Missing | N (%) | | | | | |
| Male | | | | | | |
| Female | | | | | | |
| Participant chose not to answer | | | | | | |
| Age (Mean (SD)) | XX (X.X) | | | | | |
| Age | | | | | | |
| < 18 | N (%) | | | | | |
| 18 - < 25 | | | | | | |
| 25 - < 35 | | | | | | |
| 35 - < 45 | | | | | | |
| 45 - < 55 | | | | | | |
| 55 - < 65 | | | | | | |
| 65 - < 75 | | | | | | |
| 75+ | | | | | | |
| Ethnicity | | | | | | |
| Missing | N (%) | | | | | |
| Not Hispanic or Latino | | | | | | |
| Hispanic or Latino | | | | | | |

| Table 17: Summary of | Baseline Characteristi | cs by S | tage and Tr | reatment Ar | m | |
|---|---|---|---|---|---|---|
| | | | Stage 2 | | | |
| | Stag | e 1 | Re-ran | domized | Not Re-ra | ndomized |
| Characteristic | Placebo<br>(N=) | AMC<br>(N=) | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) |
| Unknown | | | | | | |
| Participant chose not to answer | | | | | | |
| Race | | | | | | |
| Missing | N (%) | | | | | |
| American Indian or Alaska Native | | | | | | |
| Asian | | | | | | |
| Black or African American | | | | | | |
| Native Hawaiian or Pacific Islander | | | | | | |
| White | | | | | | |
| Other | | | | | | |
| Multiracial | | | | | | |
| Unknown | | | | | | |
| Participant chose not to answer | | | | | | |
| Education completed | | | | | | |
| Missing | N (%) | | | | | |
| Less than high school diploma | | | | | | |
| High school graduate | | | | | | |
| GED or equivalent | | | | | | |
| Some college, no degree | | | | | | |

| Table 17: Summary of Baseline ( | Characterist | ics by S | Stage and Ti | eatment Arı | m | |
|---|---|---|---|---|---|---|
| | | | | Stag | e 2 | |
| | Stag | je 1 | Re-ran | domized | Not Re-ra | ndomized |
| Characteristic | Placebo<br>(N=) | AMC<br>(N=) | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) |
| Associate's degree: occupational, technical, or vocational program | | | | | | |
| Associate's degree: academic program | | | | | | |
| Bachelor's degree | | | | | | |
| Master's degree | | | | | | |
| Professional school degree | | | | | | |
| Doctoral degree | | | | | | |
| Marital status | | | | | | |
| Missing | N (%) | | | | | |
| Married | | | | | | |
| Widowed | | | | | | |
| Divorced | | | | | | |
| Separated | | | | | | |
| Never married | | | | | | |
| Living with partner | | | | | | |
| Refused | | | | | | |
| Don't know | | | | | | |
| Employment | | | | | | |
| Missing | N (%) | | | | | |
| Working now | | | | | | |

| Table 17: Summary of Baseline Cl | naracterist | cs by S | tage and Ti | reatment Arı | m | |
|---|---|---|---|---|---|---|
| | | | | e 2 | | |
| | Stag | e 1 | Re-ran | domized | Not Re-randomiz | |
| Characteristic | Placebo<br>(N=) | AMC<br>(N=) | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) |
| Only temporarily laid off, sick leave, or maternity leave | | | | | | |
| Looking for work, unemployed | | | | | | |
| Retired | | | | | | |
| Disabled permanently or temporarily | | | | | | |
| Keeping house | | | | | | |
| Student | | | | | | |
| Other | | | | | | |
| Number of days of self-reported methamphetamine use in 30 days prior to informed consent | | | | | | |
| N | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Min | | | | | | |
| 25th Percentile | | | | | | |
| Median | | | | | | |
| 75th Percentile | | | | | | |
| Max | | | | | | |

| | Re-rand | domized | Not Re-rar | ndomized | |
|---|---|---|---|---|---|
| Anatomical Therapeutic Chemical Level 1/<br>Anatomical Therapeutic Chemical Level 2 | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Participants with at least one concomitant medication | | | | | |
| Gastrointestinal | N (%) | | | | |
| Acid related | N (%) | | | | |
| Antiemetics | | | | | |
| Constipation | | | | | |
| Antidiarrheal | | | | | |
| Diabetes | | | | | |
| Vitamins | | | | | |
| Mineral | | | | | |
| Other gastrointestinal | | | | | |
| Blood and Blood Forming Organs | N (%) | | | | |
| Aspirin/coumadin/heparin | N (%) | | | | |
| Anti-anemic | | | | | |
| Blood products/iv fluids | | | | | |
| Other blood and blood forming organs | | | | | |
| Cardiovascular System | N (%) | | | | |
| Antihypertensives | N (%) | | | | |
| Diuretics | | | | | |
| Beta blocking | | | | | |
| Calcium channel | | | | | |
| Lipid modifying agents | | | | | |

| | Re-rand | domized | Not Re-ran | ndomized | |
|---|---|---|---|---|---|
| Anatomical Therapeutic Chemical Level 1/<br>Anatomical Therapeutic Chemical Level 2 | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Other cardiovascular system | | | | | |
| All Skin Creams | N (%) | | | | |
| All skin creams | N (%) | | | | |
| Contraceptives/ED/Sex Hormones | N (%) | | | | |
| Contraceptives/ED/sex hormones | N (%) | | | | |
| Steroids/thyroid hormones | N (%) | | | | |
| Steroids/thyroid hormones | N (%) | | | | |
| Antibacterial/Antiviral/Antifungal/TB/Vaccines | N (%) | | | | |
| Antibacterial/antiviral/antifungal/TB/vaccines | N (%) | | | | |
| Musculoskeletal System | N (%) | | | | |
| Anti-inflammatory and antirheumatic | N (%) | | | | |
| Muscle relaxants | | | | | |
| Antigout | | | | | |
| Other musculoskeletal system | | | | | |
| Nervous System | N (%) | | | | |
| Analgesics including antipyretics | N (%) | | | | |
| Antiepileptics | | | | | |
| Anxiety/depression/sleep | | | | | |
| Other nervous system | | | | | |
| Respiratory System | N (%) | | | | |
| Nasal | N (%) | | | | |

| Table 18: Summary of Cond | comitant Medication | ns by Treat | tment Arm | ı | |
|---|---|---|---|---|---|
| | Re-rand | domized | Not Re-rar | | |
| Anatomical Therapeutic Chemical Level 1/<br>Anatomical Therapeutic Chemical Level 2 | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Throat | | | | | |
| Obstructive airway | | | | | |
| Eye and Ear Drops | N (%) | | | | |
| Eye and ear drops | N (%) | | | | |
| Various | N (%) | | | | |
| Allergens | N (%) | | | | |
| All other therapeutic products | | | | | |
| Diagnostic agents | | | | | |
| General nutrients | | | | | |
| All other non-therapeutic products | | | | | |
| Contrast media | | | | | |
| Diagnostic radiopharmaceuticals | | | | | |
| Therapeutic radiopharmaceuticals | | | | | |
| Other | N (%) | | | | |

<sup>&</sup>lt;sup>1</sup> Includes all medications taken during the safety window, which begins at the first dose date of either oral or injectable study medication, whichever comes first, and ends either 7 days after the last oral medication dose or 28 days after the last injectable medication, whichever comes last.

| Table 19: Summary of Early Medication Terminations by Site | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | SC<br>BHSPC<br>(N=) | WS<br>CODA,<br>Inc.<br>(N=) | GNY<br>SURC -<br>Columbia<br>(N=) | NS<br>Hennepin<br>Healthcare<br>(N=) | WS<br>SURU -<br>SFDPH<br>(N=) | TX UCLA<br>CBAM<br>(N=) | TX UT<br>Health<br>CNRA<br>(N=) | TX UTSW (N=) | Total<br>(N=) |
| Number of early study medication terminations <sup>1</sup> | N (%) | | | | | | | | |
| Number of participants who early terminated oral and injectable study medication | N (%) | | | | | | | | |
| Number of early oral study medication terminations | N (%) | | | | | | | | |
| Reason for early oral study medication termination | | | | | | | | | |
| Participant failed to return to site and unable to contact | N (%) | | | | | | | | |
| Participant feels treatment no longer necessary, cured | | | | | | | | | |
| Participant feels treatment no longer necessary, not working | | | | | | | | | |
| Participant interested in seeking alternate treatment | | | | | | | | | |
| Contraindicated concomitant medication | | | | | | | | | |
| Clinical deterioration: New onset of psychiatric or medical condition | | | | | | | | | |
| Clinical deterioration: Worsening of pre-existing psychiatric or medical condition | | | | | | | | | |
| Clinical deterioration: Worsening of substance use disorder | | | | | | | | | |
| Clinical deterioration: Overdose | | | | | | | | | |
| Participant became pregnant | | | | | | | | | |
| Participant withdrew consent/assent | | | | | | | | | |
| Participant reports intolerable symptoms or side effects | | | | | | | | | |
| Other | | | | | | | | | |
| Number of early injectable study medication terminations | N (%) | | | | | | | | |

| Table 19: Summary of Early Medication Terminations by Site | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | SC<br>BHSPC<br>(N=) | WS<br>CODA,<br>Inc.<br>(N=) | GNY<br>SURC -<br>Columbia<br>(N=) | NS<br>Hennepin<br>Healthcare<br>(N=) | WS<br>SURU -<br>SFDPH<br>(N=) | TX UCLA<br>CBAM<br>(N=) | TX UT<br>Health<br>CNRA<br>(N=) | TX UTSW (N=) | Total<br>(N=) |
| Reason for early injectable medication termination | | | | | | | | | |
| Participant failed to return to site and unable to contact | N (%) | | | | | | | | |
| Participant feels treatment no longer necessary, cured | | | | | | | | | |
| Participant feels treatment no longer necessary, not working | | | | | | | | | |
| Participant interested in seeking alternate treatment | | | | | | | | | |
| Contraindicated concomitant medication | | | | | | | | | |
| Clinical deterioration: New onset of psychiatric or medical condition | | | | | | | | | |
| Clinical deterioration: Worsening of pre-existing psychiatric or medical condition | | | | | | | | | |
| Clinical deterioration: Worsening of substance use disorder | | | | | | | | | |
| Clinical deterioration: Overdose | | | | | | | | | |
| Participant became pregnant | | | | | | | | | |
| Participant withdrew consent/assent | | | | | | | | | |
| Participant reports intolerable symptoms or side effects | | | | | | | | | |
| Other | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Participants who early terminated either oral or injectable study medication.

| | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
|---|---|---|---|
| Number of early study medication terminations in Stage 1 <sup>1</sup> | N (%) | | |
| Number of participants who early terminated oral and injectable study medication in Stage 1 | N (%) | | |
| Number of early oral study medication terminations in Stage 1 | N (%) | | |
| Reason for early oral study medication termination | | | |
| Participant failed to return to site and unable to contact | N (%) | | |
| Participant feels treatment no longer necessary, cured | | | |
| Participant feels treatment no longer necessary, not working | | | |
| Participant interested in seeking alternate treatment | | | |
| Contraindicated concomitant medication | | | |
| Clinical deterioration: New onset of psychiatric or medical condition | | | |
| Clinical deterioration: Worsening of pre-existing psychiatric or medical condition | | | |
| Clinical deterioration: Worsening of substance use disorder | | | |
| Clinical deterioration: Overdose | | | |
| Participant became pregnant | | | |
| Participant withdrew consent/assent | | | |
| Participant reports intolerable symptoms or side effects | | | |
| Other | | | |
| Number of early injectable study medication terminations | N (%) | | |
| Reason for early injectable study medication termination | | | |
| Participant failed to return to site and unable to contact | N (%) | | |
| Participant feels treatment no longer necessary, cured | | | |
| Participant feels treatment no longer necessary, not working | | | |
| Participant interested in seeking alternate treatment | | | |
| Contraindicated concomitant medication | | | |
| Clinical deterioration: New onset of psychiatric or medical condition | | | |
| Clinical deterioration: Worsening of pre-existing psychiatric or medical condition | | | |
| Clinical deterioration: Worsening of substance use disorder | | | |
| Clinical deterioration: Overdose | | | |
| Participant became pregnant | | | |
| Participant withdrew consent/assent | | | |
| Participant reports intolerable symptoms or side effects | | | |

<sup>&</sup>lt;sup>1</sup> Participants who early terminated either oral study medication before the date of re-randomization or Day 43 for non-re-randomized participants, or early terminated injectable study medication and received no injections or only injection #1.

| | Re-randomized | | Not Re-rar | | |
|---|---|---|---|---|---|
| | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Number of early study medication terminations in Stage 2 <sup>1</sup> | N (%) | | | | |
| Number of participants who early terminated oral and injectable study medication in Stage 2 | N (%) | | | | |
| Number of early oral study medication terminations in Stage 2 | N (%) | | | | |
| Reason for early oral study medication termination | | | | | |
| Participant failed to return to site and unable to contact | N (%) | | | | |
| Participant feels treatment no longer necessary, cured | | | | | |
| Participant feels treatment no longer necessary, not working | | | | | |
| Participant interested in seeking alternate treatment | | | | | |
| Contraindicated concomitant medication | | | | | |
| Clinical deterioration: New onset of psychiatric or medical condition | | | | | |
| Clinical deterioration: Worsening of pre-existing psychiatric or medical condition | | | | | |
| Clinical deterioration: Worsening of substance use disorder | | | | | |
| Clinical deterioration: Overdose | | | | | |
| Participant became pregnant | | | | | |
| Participant withdrew consent/assent | | | | | |
| Participant reports intolerable symptoms or side effects | | | | | |
| Other | | | | | |
| Number of early injectable study medication terminations | N (%) | | | | |
| Reason for early injectable study medication termination | | | | | |
| Participant failed to return to site and unable to contact | N (%) | | | | |
| Participant feels treatment no longer necessary, cured | | | | | |
| Participant feels treatment no longer necessary, not working | | | | | |
| Participant interested in seeking alternate treatment | | | | | |
| Contraindicated concomitant medication | | | | | |
| Clinical deterioration: New onset of psychiatric or medical condition | | | | | |
| Clinical deterioration: Worsening of pre-existing psychiatric or medical condition | | | | | |
| Clinical deterioration: Worsening of substance use disorder | | | | | |
| Clinical deterioration: Overdose | | | | | |
| Participant became pregnant | | | | | |
| Participant withdrew consent/assent | | | | | |
| Participant reports intolerable symptoms or side effects | | | | | |
| Other | | | | | |

<sup>&</sup>lt;sup>1</sup> Participants who early terminated either oral study medication on or after the date of re-randomization or Day 43 for non-re-randomized participants, or early terminated injectable study medication after last receiving injection #2 or #3.

| | Table 22: Summary of Treatment Exposure by Site | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Tablets <sup>1</sup> | | | Inje | | Overall<br>Treatment<br>Exposure <sup>2</sup> | |
| Site | Participants<br>Randomized | Taken | Expected | % | Administered | Expected | % | % |
| SC BHSPC | N | N | N | % | N | N | % | % |
| WS CODA, Inc. | | | | | | | | |
| GNY SURC - Columbia | | | | | | | | |
| NS Hennepin Healthcare | | | | | | | | |
| WS SURU - SFDPH | | | | | | | | |
| TX UCLA CBAM | | | | | | | | |
| TX UT Health CNRA | | | | | | | | |
| TX UTSW | | | | | | | | |
| Total | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Three tablets per day are expected during the 12-week treatment period.

<sup>&</sup>lt;sup>2</sup> Four injections are expected during the 12-week treatment period.

<sup>&</sup>lt;sup>3</sup> Overall treatment exposure percentage is an average of the percentage for tablets and percentage for injections. This percentage represents medication adherence across all treatment groups (i.e., Placebo, AMC, Placebo, Placebo, placebo/AMC).

| Table | 23: Summ | ary of Treatment I | Exposure | by Site, | Stage and | Treatmen | t Arm | |
|---|---|---|---|---|---|---|---|---|
| | | | | e 2 | | | | |
| | | | Stag | e 1 | Re-rand | domized | Not Re-ra | ndomized |
| Site | Treatment | Exposure | Placebo<br>(N=) | AMC<br>(N=) | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) |
| SC BHSPC | Tablets <sup>1</sup> | Number Taken | N | | | | | |
| | | Number Expected | N | | | | | |
| | | Percent Taken | % | | | | | |
| | Injections <sup>2</sup> | Number Administered | N | | | | | |
| | | Number Expected | N | | | | | |
| | | Percent Administered | % | | | | | |
| | Overall <sup>3</sup> | Treatment Exposure | % | | | | | |
| WS CODA, Inc. | Tablets <sup>1</sup> | Number Taken | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Taken | | | | | | |
| | Injections <sup>2</sup> | Number Administered | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Administered | | | | | | |
| | Overall <sup>3</sup> | Treatment Exposure | | | | | | |
| GNY SURC - Columbia | Tablets <sup>1</sup> | Number Taken | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Taken | | | | | | |
| | Injections <sup>2</sup> | Number Administered | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Administered | | | | | | |
| | Overall <sup>3</sup> | Treatment Exposure | | | | | | |
| NS Hennepin Healthcare | Tablets <sup>1</sup> | Number Taken | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Taken | | | | | | |
| | Injections <sup>2</sup> | Number Administered | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Administered | | | | | | |
| | Overall <sup>3</sup> | Treatment Exposure | | | | | | |

| | | | | | | Stag | e 2 | |
|---|---|---|---|---|---|---|---|---|
| | | | Stag | e 1 | Re-rand | domized | Not Re-randomized | |
| Site | Treatment | Exposure | Placebo<br>(N=) | AMC<br>(N=) | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) |
| WS SURU - SFDPH | Tablets <sup>1</sup> | Number Taken | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Taken | | | | | | |
| | Injections <sup>2</sup> | Number Administered | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Administered | | | | | | |
| | Overall <sup>3</sup> | Treatment Exposure | | | | | | |
| TX UCLA CBAM | Tablets <sup>1</sup> | Number Taken | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Taken | | | | | | |
| | Injections <sup>2</sup> | Number Administered | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Administered | | | | | | |
| | Overall <sup>3</sup> | Treatment Exposure | | | | | | |
| TX UT Health CNRA | Tablets <sup>1</sup> | Number Taken | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Taken | | | | | | |
| | Injections <sup>2</sup> | Number Administered | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Administered | | | | | | |
| | Overall <sup>3</sup> | Treatment Exposure | | | | | | |
| Total | Tablets <sup>1</sup> | Number Taken | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Taken | | | | | | |
| | Injections <sup>2</sup> | Number Administered | | | | | | |
| | | Number Expected | | | | | | |
| | | Percent Administered | | | | | | |
| | Overall <sup>3</sup> | Treatment Exposure | 1 | | 1 | | 1 | |

<sup>&</sup>lt;sup>1</sup> Three tablets per day are expected during Stage 1 (Weeks 1-6) and Stage 2 (Weeks 7-12).

<sup>&</sup>lt;sup>2</sup> Two injections are expected in each stage.

<sup>&</sup>lt;sup>3</sup> Overall treatment exposure percentage is an average of the percentage for tablets and percentage for injections.

| | Table 24: Summary of Injections by Site | | | | |
|---|---|---|---|---|---|
| Site | Participants<br>Randomized | Participants<br>Who<br>Received<br>Injection #1 | Participants<br>Who<br>Received<br>Injection #2 | Participants<br>Who<br>Received<br>Injection #3 | Participants<br>Who<br>Received<br>Injection #4 |
| SC BHSPC | N | N (%) | N (%) | N (%) | N (%) |
| WS CODA, Inc. | | | | | |
| GNY SURC - Columbia | | | | | |
| NS Hennepin Healthcare | | | | | |
| WS SURU - SFDPH | | | | | |
| TX UCLA CBAM | | | | | |
| TX UT Health CNRA | | | | | |
| TX UTSW | | | | | |
| Total | | | | | |

| Table 25: Summary of Injections by Stage and Treatment Arm | | | | | | | | | |
|---|---|---|---|---|---|---|--|--|--|
| | | | | Stag | e 2 | | | | |
| | Stag | je 1 | Re-rand | domized | Not Re-ra | ndomized | | | |
| | Placebo<br>(N=) | AMC<br>(N=) | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | | | |
| Participants who received injection #1 | N (%) | | | | | | | | |
| Participants who received injection #2 | N (%) | | | | | | | | |
| Participants who received injection #3 | | | N (%) | | | | | | |
| Participants who received injection #4 | | | N (%) | | | | | | |
| Table 26: Summa | ry of Oral Medi<br>AMC Parti | | evels by Stage | | | | |
|---|---|---|---|---|--|--|--|
| | Stage 1 | | Stage 2 | | | | |
| | | Re-randomized | Not<br>Re-randomized | | | | |
| | AMC<br>(N=) | Placebo/<br>AMC<br>(N=) | AMC<br>(N=) | Total<br>(N=) | | | |
| Bupropion adherence <sup>1</sup> | | | | | | | |
| Visit 0401 | n/N (%) | | | | | | |
| Visit 0701 | | | | | | | |
| Visit 1001 | | | | | | | |
| Visit 1201 | | | | | | | |
| Hydroxybupropion adherence <sup>2</sup> | | | | | | | |
| Visit 0401 | n/N (%) | | | | | | |
| Visit 0701 | | | | | | | |
| Visit 1001 | | | | | | | |
| Visit 1201 | | | | | | | |

<sup>&</sup>lt;sup>1</sup> A participant is considered adherent if bupropion blood level is greater than 0.500 ng/mL.

<sup>&</sup>lt;sup>2</sup> A participant is considered adherent if hydroxybupropion blood level is greater than 1.00 ng/mL.

| Table 27: Summary of Primary Outcome Availability by Stage and Treatment Arm ITT Population | | | | | |
|---|---|---|---|---|---|
| | | | Re-rand | lomized | |
| | Stag<br>(Weeks | | | | |
| | Placebo<br>(N=) | AMC<br>(N=) | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Total<br>(N=) |
| Number of UDS methamphetamine results collected <sup>1</sup> | N | | | | |
| Number of UDS expected <sup>2</sup> | N | | | | |
| Percentage of expected UDS methamphetamine results collected | % | | | | |

<sup>&</sup>lt;sup>1</sup> Number of UDS with methamphetamine results collected in Weeks 5 and 6 in Stage 1 and Weeks 11 and 12 in Stage 2

<sup>&</sup>lt;sup>2</sup> Two UDS are expected per participant each week.

| | Table 28: Summary of Primary Outcome Analysis by Stage and Treatment Arm ITT Population | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Design Par | Design Parameters Stage 1 Stage 2 Results | | | | | | | | | | | |
| Random-<br>ization<br>fraction a | Weight w | N | Placebo<br>Responder<br>Rate <i>q1</i> | AMC<br>Responder<br>Rate <i>p1</i> | Rate of<br>Continuation<br>into Stage 2<br>among<br>Placebo Non-<br>responders s | Placebo<br>Responder<br>Rate <i>q2</i> | AMC<br>Responder<br>Rate <i>p2</i> | Treatment<br>Effect h | Standard<br>Error of h | Wald<br>Type<br>Test<br>Statistic<br>Z | p-value <sup>1</sup> | 95% Lower<br>Confidence<br>Limit |
| 0.37 | 0.43 N X/X (X.X%) X/X (X.X%) X.XXXX N X/X (X.X%) X/X (X.X%) X.XXXX X.XXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXX X.XXXX X.XXX X.XX X.XXX X.XX X.XXX X.XX X.XX X.XXX X.X | | | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> The p-value was calculated adjusting for interim efficacy analysis.

Figure 7: Methamphetamine Negative UDS Results by Stage and Treatment Arm ITT Population



| | Γable 29: Summary of Pri | • | ne Sensitivi<br>ITT Populat | • | s by Stage a | nd Treatmer | nt Arm | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Stage 1 | | | Stage 2 | | Resi | ults |
| Method | Results | Number<br>Randomized | Placebo<br>Responder<br>Rate <i>q1</i> | AMC<br>Responder<br>Rate <i>p1</i> | Number Re-<br>randomized | Placebo<br>Responder<br>Rate <i>q2</i> | AMC<br>Responder<br>Rate <i>p2</i> | Treatment<br>Effect h | Standard<br>Error of h |
| Protocol defined primary outcome | Primary outcome | N | X/X (X.X%) | X/X (X.X%) | N | X/X (X.X%) | X/X (X.X%) | X.XXXX | X.XXXX |
| Imputation of missing UDS | Missing UDS imputed as negative | | | | | | | | |
| | Missing UDS imputed as positive | | | | | | | | |
| | Complete cases <sup>1</sup> | | | | | | | | |
| Using weight w=0.5 | Adjusted primary outcome | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Includes participants with all four UDS collected in the stage.

| | | | | | Re-randomized | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | tage 1<br>eeks 5-6) | | Stage 2<br>(Weeks 11-12) | | | | |
| Site | N | Number of UDS methamphetamine results collected | Number of<br>UDS<br>expected <sup>1</sup> | Percentage of expected UDS methamphetamine results collected | N | Number of UDS methamphetamine results collected | Number of<br>UDS<br>expected <sup>1</sup> | Percentage of expected UDS methamphetamine results collected | Total |
| SC BHSPC | XX | XXX | XXX | XX.X% | XX | XXX | XXX | XX.X% | XX.X% |
| WS CODA, Inc. | | | | | | | | | |
| GNY SURC - Columbia | | | | | | | | | |
| NS Hennepin Healthcare | | | | | | | | | |
| WS SURU - SFDPH | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | |
| TX UTSW | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup>Two UDS are expected per participant in Weeks 5, 6, 11, and 12.

| | Table 31: | Summary o | | Outcome by Si<br>IT Population | te, Stage, a | and Treatm | ent Arm | | |
|---|---|---|---|---|---|---|---|---|---|
| | Stage 1 | | | Stage 2 | | | Results <sup>1</sup> | | |
| Site | Number<br>Randomized | Placebo<br>Responder<br>Rate <i>q1</i> | AMC<br>Responder<br>Rate <i>p1</i> | Number<br>Re-randomized | Placebo<br>Responder<br>Rate q2 | AMC<br>Responder<br>Rate p2 | Treatment<br>Effect h | Standard<br>Error of h | p-value |
| SC BHSPC | N | X/X (X.X%) | X/X (X.X%) | N | X/X (X.X%) | X/X (X.X%) | X.XXXX | X.XXXX | X.XXXX |
| WS CODA, Inc. | | | | | | | | | |
| GNY SURC - Columbia | | | | | | | | | |
| NS Hennepin Healthcare | | | | | | | | | |
| WS SURU - SFDPH | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | |
| TX UTSW | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Results are obtained from the generalized linear mixed effects model.

| | Table 32: Summary of Primary Outcome by Sex, Stage, and Treatment Arm ITT Population | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Stage 1 Stage 2 Results <sup>1</sup> | | | | | | | | |
| Subgroup | Number<br>Randomized | Placebo<br>Responder<br>Rate <i>q1</i> | AMC<br>Responder<br>Rate <i>p1</i> | Number<br>Re-randomized | Placebo<br>Responder<br>Rate <i>q2</i> | AMC<br>Responder<br>Rate <i>p2</i> | Treatment<br>Effect h | Standard<br>Error of <i>h</i> | p-value |
| Male | N | X/X (X.X%) | X/X (X.X%) | N | X/X (X.X%) | X/X (X.X%) | X.XXXX | X.XXXX | X.XXXX |
| Female | N | X/X (X.X%) | X/X (X.X%) | N | X/X (X.X%) | X/X (X.X%) | X.XXXX | X.XXXX | |

<sup>&</sup>lt;sup>1</sup> Results are obtained from a generalized linear mixed effects model.

| Table 33: Summary of Primary Outcome by Race, Stage, and Treatment Arm ITT Population | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Stage 1 Stage 2 Results <sup>1</sup> | | | | | | | | | |
| Subgroup | Number<br>Randomized | Placebo<br>Responder<br>Rate <i>q1</i> | AMC<br>Responder<br>Rate <i>p1</i> | Number<br>Re-randomized | Placebo<br>Responder<br>Rate <i>q2</i> | AMC<br>Responder<br>Rate <i>p2</i> | Treatment<br>Effect h | Standard<br>Error of <i>h</i> | |
| Black or African American | N | X/X (X.X%) | X/X (X.X%) | N | X/X (X.X%) | X/X (X.X%) | X.XXXX | X.XXXX | X.XXXX |
| White | N | X/X (X.X%) | X/X (X.X%) | N | X/X (X.X%) | X/X (X.X%) | X.XXXX | X.XXXX | |
| Other <sup>2</sup> | her <sup>2</sup> N X/X (X.X%) X/X (X.X%) N X/X (X.X%) X/X (X.X%) X.XXXX X.XXXX | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Results are obtained from a generalized linear mixed effects model.

| Table 34: Summary of Primary Outcome by Ethnicity, Stage, and Treatment Arm ITT Population | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Stage 1 Stage 2 Results <sup>1</sup> | | | | | | | | | |
| Subgroup | Number<br>Randomized | Placebo<br>Responder<br>Rate <i>q1</i> | AMC<br>Responder<br>Rate <i>p1</i> | Number<br>Re-randomized | Placebo<br>Responder<br>Rate <i>q2</i> | AMC<br>Responder<br>Rate <i>p2</i> | Treatment<br>Effect h | Standard<br>Error of h | p-value |
| Hispanic or Latino | spanic or Latino N X/X (X.X%) X/X (X.X%) N X/X (X.X%) X/X (X.X%) X/X (X.X%) X/X (X.XXX) X.XXXXX X.XXXXX | | | | | | | | |
| Not Hispanic or Latino/Other <sup>2</sup> N X/X (X.X%) X/X (X.X%) N X/X (X.X%) X/X (X.X%) X.XXXX X.XXXX | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Results are obtained from a generalized linear mixed effects model.

<sup>&</sup>lt;sup>2</sup> Includes American Indian or Alaska Native, Asian, Native Hawaiian or Pacific Islander, Multiracial, Other, Don't Know, and Refused to Answer.

<sup>&</sup>lt;sup>2</sup> Includes Not Hispanic or Latino, Don't Know, and Refused to Answer.

| | Table 35: Summary of Primary Outcome by Age, Stage, and Treatment Arm ITT Population | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Stage 1 Stage 2 Results <sup>1</sup> | | | | | | | | |
| Subgroup | Number<br>Randomized | Placebo<br>Responder<br>Rate <i>q1</i> | AMC<br>Responder<br>Rate <i>p1</i> | Number<br>Re-randomized | Placebo<br>Responder<br>Rate <i>q2</i> | AMC<br>Responder<br>Rate <i>p2</i> | Treatment<br>Effect h | Standard<br>Error of h | p-value |
| ≤ 40 years | N | N X/X (X.X%) X/X (X.X%) N X/X (X.X%) X/X (X.X%) X.XXXX X.XXXX | | | | | | | |
| > 40 years | N | N X/X (X.X%) X/X (X.X%) N X/X (X.X%) X/X (X.X%) X.XXXX X.XXXX | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Results are obtained from a generalized linear mixed effects model.

| Table 36: Primary Outcome Covariate Adjusted Analysis Results <sup>1</sup> ITT Population | | | |
|---|---|---|---|
| Model Results | Treatment<br>Effect <i>h</i> | Standard<br>Error of <i>h</i> | p-value |
| Treatment Effect | X.XXXX | X.XXXX | X.XXXX |
| Other Covariates in the Model | | | |
| Site | | | X.XXXX |
| Age at onset of methamphetamine use | | | X.XXXX |
| Baseline number of methamphetamine use days self-reported | | | X.XXXX |
| Baseline IV methamphetamine use self-reported | | | X.XXXX |
| Number of DSM-5 criteria met during screening | | | X.XXXX |
| Baseline number of days of cigarette or e-cigarette use self-reported | | | X.XXXX |
| Baseline Treatment Effectiveness Assessment Score | | | X.XXXX |
| Baseline average Visual Analog Craving Scale Score | | | X.XXXX |

<sup>&</sup>lt;sup>1</sup>Results are obtained from a generalized linear mixed effects model.

| Table | 37: Summa | | Availability <sup>1</sup><br>lomized Pop | | ınd Treatme | ent Arm |
|---|---|---|---|---|---|---|
| | | | | Stag | је 2 | |
| | Stag | ge 1 | Re-rand | lomized | Not Re-rai | ndomized |
| Weeks | Placebo<br>(N=) | AMC<br>(N=) | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) |
| 1-2 | n/N (%) | | | | | |
| 3-4 | | | | | | |
| 5-6 <sup>2</sup> | | | | | | |
| 7-8 | | | | | | |
| 9-10 | | | | | | |
| 11-12 <sup>2</sup> | | | | | | |
| 13³ | | | | | | |
| 16³ | | | | | | |

<sup>&</sup>lt;sup>1</sup> UDS Availability is presented as number of collected UDS over number of expected UDS. Two UDS per participant are expected each week, with the exception of one UDS expected during Week 1. A UDS is considered collected if the UDS has a methamphetamine result.

<sup>&</sup>lt;sup>2</sup>Weeks 5-6 and 11-12 are the primary outcome evaluation period.

<sup>&</sup>lt;sup>3</sup> Week 13 and Week 16 occur during the Follow-up Period. One UDS per participant per visit is expected at Week 13 and at Week 16.

Table 38: Summary of Methamphetamine Negative UDS Results by Treatment Arm in Stage 1 Randomized Population

| Visit | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
|-------|-----------------|-------------|---------------|
| 0101 | n/N (%) | | |
| 0102 | | | |
| 0201 | | | |
| 0202 | | | |
| 0301 | | | |
| 0302 | | | |
| 0401 | | | |
| 0402 | | | |
| 0501 | | | |
| 0502 | | | |
| 0601 | | | |
| 0602 | | | |

# Table 39: Summary of Methamphetamine Negative UDS Results by Treatment Arm in Stage 2 Randomized Population

| | 1 | | 1 | | |
|---|---|---|---|---|---|
| | Re-rand | lomized | Not Re-ra | ndomized | |
| Visit | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| 0701 | n/N (%) | | | | |
| 0702 | | | | | |
| 0801 | | | | | |
| 0802 | | | | | |
| 0901 | | | | | |
| 0902 | | | | | |
| 1001 | | | | | |
| 1002 | | | | | |
| 1101 | | | | | |
| 1102 | | | | | |
| 1201 | | | | | |
| 1202 | | | | | |

Table 40: Summary of Methamphetamine Negative UDS Results by Treatment Arm in Follow-up Period Randomized Population

| | Re-randomized Not Re-randomized | | | | |
|---|---|---|---|---|---|
| Visit | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| 1301 | n/N (%) | | | | |
| 1601 | | | | | |

| | Table 41: Summary of Pri | imary | | ensitivity An<br>zed Populati | | y Stage and | Treatment A | rm | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Stage 1 Stage 2 | | | | | | | | |
| | | | | | | Re-randomiz | ed | | Not Re-rando | mized |
| Method | Results | N | Placebo<br>Responder<br>Rate <i>q1</i> | AMC<br>Responder<br>Rate <i>p1</i> | N | Placebo/<br>Placebo<br>Responder<br>Rate <i>q2</i> | Placebo/<br>AMC<br>Responder<br>Rate <i>p2</i> | N | Placebo<br>Responder<br>Rate | AMC<br>Responder<br>Rate |
| Protocol defined primary outcome | Primary outcome | N | X/X (X.X%) | X/X (X.X%) | N | X/X (X.X%) | X/X (X.X%) | N | X/X (X.X%) | X/X (X.X%) |
| Imputation of missing UDS | Missing UDS imputed as negative | | | | | | | | | |
| | Missing UDS imputed as positive | | | | | | | | | |
| | Complete cases <sup>1</sup> | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Includes participants with all four UDS collected in the stage.

Figure 8: Methamphetamine Negative UDS Results by Stage and Treatment Arm Randomized Population



| Table 42: Summary of Primary Outcome by Stage and Treatment Arm Per Protocol Populations | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Stage 1 Stage 2 Result | | | | | | | | ults |
| Per Protocol Population | Number<br>Randomized | Placebo<br>Responder<br>Rate <i>q1</i> | AMC<br>Responder<br>Rate <i>p1</i> | Number<br>Re-randomized | Placebo<br>Responder<br>Rate <i>q2</i> | AMC<br>Responder<br>Rate <i>p2</i> | Treatment<br>Effect h | Standard<br>Error of h |
| Definition 1 | N | X.X (X.X%) | X.X (X.X%) | N | X.X (X.X%) | X.X (X.X%) | X.XXXX | X.XXXX |
| Definition 2 | N | X.X (X.X%) | X.X (X.X%) | N | X.X (X.X%) | X.X (X.X%) | X.XXXX | X.XXXX |
| Definition 4 | N | | X.X (X.X%) | N | | X.X (X.X%) | | |

| Table 43: Summary of Treatment Emergent Adverse Events | ents by Tr | eatment | Arm in |
|---|---|---|---|
| | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Number of participants with treatment emergent adverse events in Stage 1 <sup>1</sup> | N (%) | | |
| Number of treatment emergent adverse events | N | | |
| Severity of adverse event | | | |
| Missing | N (%) | | |
| Grade 1 - Mild | | | |
| Grade 2 - Moderate | | | |
| Grade 3 - Severe | | | |
| Relationship of treatment emergent adverse event to oral study medication | | | |
| Missing | N (%) | | |
| No | | | |
| Yes | | | |
| Relationship of treatment emergent adverse event to injectable study medication | | | |
| Missing | N (%) | | |
| No | | | |
| Yes | | | |

<sup>&</sup>lt;sup>1</sup> Stage 1 AEs include adverse events occurring before the date of re-randomization for re-randomized participants and in Weeks 1-6 for non-re-randomized participants.

| | Re-rand | domized | Not Re-rai | | |
|---|---|---|---|---|---|
| | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Number of participants with treatment emergent adverse events in Stage 2 <sup>1</sup> | N (%) | | | | |
| Number of treatment emergent adverse events | N | | | | |
| Severity of adverse event | | | | | |
| Missing | N (%) | | | | |
| Grade 1 - Mild | | | | | |
| Grade 2 - Moderate | | | | | |
| Grade 3 - Severe | | | | | |
| Relationship of treatment emergent adverse event to oral study medication | | | | | |
| No | N (%) | | | | |
| Yes | | | | | |
| Relationship of treatment emergent adverse event to injectable study medication | | | | | |
| No | N (%) | | | | |
| Yes | | | | | |

Yes

1 Stage 2 AEs include adverse events occurring on or after the date of re-randomization for re-randomized participants and in Weeks 7 or greater for non-re-randomized participants.

| System Organ Class/<br>Preferred Term (MedDRA v22.0) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
|---|---|---|---|
| Participants with at least one adverse event in Stage 1 <sup>1</sup> | N (%) | | |
| Gastrointestinal disorders | N (%) | | |
| Nausea | N (%) | | |
| Diarrhoea | | | |
| Constipation | | | |
| Vomiting | | | |
| Dry mouth | | | |
| Toothache | | | |
| Abdominal discomfort | | | |
| Abdominal pain upper | | | |
| Abdominal pain | | | |
| Dyspepsia | | | |
| Chapped lips | | | |
| Breath odour | | | |
| Abdominal pain lower | | | |
| Vomiting projectile | | | |
| Stomatitis | | | |
| Rectal haemorrhage | | | |
| Abdominal distension | | | |
| Pancreatitis | | | |
| Oral disorder | | | |
| Melaena | | | |
| Loose tooth | | | |
| Gastrooesophageal reflux disease | | | |
| Gastrointestinal pain | | | |
| Gastritis | | | |
| Food poisoning | | | |
| Psychiatric disorders | N (%) | | |
| Anxiety | N (%) | | |
| Insomnia | | | |
| Irritability | | | |
| Affect lability | | | |
| Abnormal dreams | | | |
| Depression | | | |

| System Organ Class/<br>Preferred Term (MedDRA v22.0) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
|---|---|---|---|
| Depressed mood | | | |
| Libido decreased | | | |
| Nervous system disorders | N (%) | | |
| Headache | N (%) | | |
| Dizziness | | | |
| Somnolence | | | |
| Lethargy | | | |
| Tremor | | | |
| Dysgeusia | | | |
| Cognitive disorder | | | |
| Hypersomnia | | | |
| Head discomfort | | | |
| Loss of consciousness | | | |
| Hypoaesthesia | | | |
| Disturbance in attention | | | |
| Depressed level of consciousness | | | |
| Syncope | | | |
| Restless legs syndrome | | | |
| Parosmia | | | |
| Nerve compression | | | |
| Migraine | | | |
| Infections and infestations | N (%) | | |
| Upper respiratory tract infection | N (%) | | |
| Nasopharyngitis | | | |
| Cellulitis | | | |
| Gonorrhoea | | | |
| Gastroenteritis | | | |
| Urinary tract infection | | | |
| Syphilis | | | |
| Abscess | | | |
| Viral infection | | | |
| Abscess limb | | | |
| Pharyngitis | | | |
| Influenza | | | |

| System Organ Class/<br>Preferred Term (MedDRA v22.0) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
|---|---|---|---|
| Gastroenteritis viral | , , | . , | , , |
| Furuncle | | | |
| Ear infection | | | |
| Cystitis | | | |
| General disorders and administration site conditions | N (%) | | |
| Fatigue | N (%) | | |
| Pain | | | |
| Feeling jittery | | | |
| Injury, poisoning and procedural complications | N (%) | | |
| Laceration | N (%) | | |
| Contusion | | | |
| Skin abrasion | | | |
| Thermal burn | | | |
| Road traffic accident | | | |
| Ligament sprain | | | |
| Injection site pain | | | |
| Skin and subcutaneous tissue disorders | N (%) | | |
| Hyperhidrosis | N (%) | | |
| Rash | | | |
| Acne | | | |
| Ecchymosis | | | |
| Eczema | | | |
| Blister | | | |
| Laceration | | | |
| Erythema | | | |
| Musculoskeletal and connective tissue disorders | N (%) | | |
| Myalgia | N (%) | | |
| Arthralgia | | | |
| Back pain | | | |

<sup>&</sup>lt;sup>1</sup> Stage 1 AEs include adverse events occurring before the date of re-randomization for re-randomized participants and in Weeks 1-6 for non-re-randomized participants.

# Table 46: Summary of Treatment Emergent MedDRA Coded Adverse Events by Treatment Arm in Stage 2

| | Re-rand | lomized | Not Re-rar | | |
|---|---|---|---|---|---|
| System Organ Class/<br>Preferred Term (MedDRA v22.0) | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Participants with at least one adverse event in Stage 2 <sup>1</sup> | N (%) | | | | |
| Infections and infestations | N (%) | | | | |
| Nasopharyngitis | N (%) | | | | |
| Upper respiratory tract infection | | | | | |
| Cellulitis | | | | | |
| Paronychia | | | | | |
| Oral herpes | | | | | |
| Abscess | | | | | |
| Viral infection | | | | | |
| Pneumonia | | | | | |
| Influenza | | | | | |
| Herpes virus infection | | | | | |
| Gastroenteritis viral | | | | | |
| Epididymitis | | | | | |
| Chlamydial infection | | | | | |
| Breast abscess | | | | | |
| Body tinea | | | | | |
| Urosepsis | | | | | |
| Urinary tract infection | | | | | |
| Appendicitis | | | | | |
| Tooth abscess | | | | | |
| Tinea infection | | | | | |
| Syphilis | | | | | |
| Pharyngitis | | | | | |
| Infectious mononucleosis | | | | | |
| Gastrointestinal disorders | N (%) | | | | |
| Nausea | N (%) | | | | |
| Vomiting | | | | | |
| Abdominal pain upper | | | | | |
| Diarrhoea | | | | | |
| Constipation | | | | | |
| Dyspepsia | | | | | |
| Abdominal discomfort | | | | | |

### Table 46: Summary of Treatment Emergent MedDRA Coded Adverse Events by Treatment Arm in Stage 2

| | Re-rand | domized | Not Re-ran | domized | |
|---|---|---|---|---|---|
| System Organ Class/<br>Preferred Term (MedDRA v22.0) | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Toothache | | | | | |
| Gastritis | | | | | |
| Flatulence | | | | | |
| Dry mouth | | | | | |
| Abdominal pain | | | | | |
| Glossodynia | | | | | |
| General disorders and administration site conditions | N (%) | | | | |
| Fatigue | N (%) | | | | |
| Pain | | | | | |
| Influenza like illness | | | | | |
| Chest pain | | | | | |
| Pyrexia | | | | | |
| Asthenia | | | | | |
| Injection site swelling | | | | | |
| Injection site haematoma | | | | | |
| Injection site discomfort | | | | | |
| Drug withdrawal syndrome | | | | | |
| Vessel puncture site bruise | | | | | |
| Peripheral swelling | | | | | |
| njury, poisoning and procedural complications | N (%) | | | | |
| Laceration | N (%) | | | | |
| Joint injury | | | | | |
| Arthropod bite | | | | | |
| Muscle strain | | | | | |
| Eye injury | | | | | |
| Contusion | | | | | |
| Thermal burn | | | | | |
| Road traffic accident | | | | | |
| Procedural nausea | | | | | |
| Limb injury | | | | | |
| Ligament sprain | | | | | |
| Skin abrasion | | | | | |
| Nervous system disorders | N (%) | | | | |

### Table 46: Summary of Treatment Emergent MedDRA Coded Adverse Events by Treatment Arm in Stage 2

| | Re-rand | domized | Not Re-rar | | |
|---|---|---|---|---|---|
| System Organ Class/<br>Preferred Term (MedDRA v22.0) | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Headache | N (%) | | | | |
| Dizziness | | | | | |
| Dysgeusia | | | | | |
| Tremor | | | | | |
| Nerve compression | | | | | |
| Migraine | | | | | |
| Psychiatric disorders | N (%) | | | | |
| Depression | N (%) | | | | |
| Anxiety | | | | | |
| Paranoia | | | | | |
| Insomnia | | | | | |
| Homicidal ideation | | | | | |
| Hallucination | | | | | |
| Feeling guilty | | | | | |
| Disorientation | | | | | |
| Anhedonia | | | | | |
| Musculoskeletal and connective tissue disorders | N (%) | | | | |
| Myalgia | N (%) | | | | |
| Pain in extremity | | | | | |
| Back pain | | | | | |
| Musculoskeletal pain | | | | | |
| Neck pain | | | | | |
| Musculoskeletal chest pain | | | | | |
| Muscular weakness | | | | | |
| Joint stiffness | | | | | |
| Arthralgia | | | | | |
| Pain in jaw | | | | | |

<sup>&</sup>lt;sup>1</sup> Stage 2 AEs include adverse events occurring on or after the date of re-randomization for re-randomized participants and in Weeks 7 or greater for non-re-randomized participants.

## Listing 1: Treatment Emergent Adverse Events by Treatment Arm Treatment Arm = Placebo

| | | | | | | | | | | | MedDR | A v22.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Participant ID | Random-<br>ization<br>Date | Onset<br>Date | AE<br>Description | Severity<br>of AE | Related-<br>ness to<br>Oral<br>Study<br>Drug | Related-<br>ness to<br>Injectable<br>Study<br>Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| SC BHSPC | | | | | | | | | | | | |
| WS CODA,<br>Inc. | | | | | | | | | | | | |
| GNY SURC -<br>Columbia | | | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | | | |
| WS SURU -<br>SFDPH | | | | | | | | | | | | |
| TX UCLA<br>CBAM | | | | | | | | | | | | |
| TX UT Health<br>CNRA | | | | | | | | | | | | |
| TX UTSW | | | | | | | | | | | | |

## Listing 1: Treatment Emergent Adverse Events by Treatment Arm Treatment Arm = Placebo/Placebo

| | | | | | | | | | | | | MedDR | A v22.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Participant ID | Random-<br>ization<br>Date | Re-ran-<br>domi-<br>-zation<br>Date | Onset<br>Date | AE<br>Description | Severity<br>of AE | Related-<br>ness to<br>Oral<br>Study<br>Drug | Related-<br>ness to<br>Injectable<br>Study<br>Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associ-<br>ated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| SC BHSPC | | | | | | | | | | | | | |
| WS CODA,<br>Inc. | | | | | | | | | | | | | |
| GNY SURC -<br>Columbia | | | | | | | | | | | | | |
| NS<br>Hennepin<br>Healthcare | | | | | | | | | | | | | |
| WS SURU -<br>SFDPH | | | | | | | | | | | | | |
| TX UCLA<br>CBAM | | | | | | | | | | | | | |
| TX UT<br>Health<br>CNRA | | | | | | | | | | | | | |
| TX UTSW | | | | | | | | | | | | | |

## Listing 1: Treatment Emergent Adverse Events by Treatment Arm Treatment Arm = Placebo/AMC

MedDRA v22.0 and higher Related-Relatedness to ΑE Re-ranness to domi-Oral Injectable Resolu-**System** Random-Associ-Preferred Onset ΑE Severity Study Órgan ization zation Study tion ated Outcome Class With Site Participant ID Date Date Date Description of AE Drug Drug Date Term SC BHSPC WS CODA, Inc. GNY SURC -Columbia NS Hennepin Healthcare WS SURU -SFDPH TX UCLA CBAM TX UT Health CNRA

SAEs are highlighted in gray.

TX UTSW

## Listing 1: Treatment Emergent Adverse Events by Treatment Arm Treatment Arm = AMC

| | | | | | | | | | | | | v22.0 and<br>her |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Participant ID | Random-<br>ization<br>Date | Onset<br>Date | AE<br>Description | Severity<br>of AE | Related<br>-ness<br>to Oral<br>Study<br>Drug | Related<br>-ness to<br>Injectable<br>Study<br>Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| SC BHSPC | | | | | | | | | | | | |
| WS CODA,<br>Inc. | | | | | | | | | | | | |
| GNY SURC -<br>Columbia | | | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | | | |
| WS SURU -<br>SFDPH | | | | | | | | | | | | |
| TX UCLA<br>CBAM | | | | | | | | | | | | |
| TX UT Health<br>CNRA | | | | | | | | | | | | |
| TX UTSW | | | | | | | | | | | | |

## Listing 2: Non-Treatment Emergent Adverse Events in Randomized Participants by Treatment Arm Treatment Arm = Placebo

| | | | | | | | | | | | MedDR | A v22.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Participant ID | Random-<br>ization<br>Date | Onset<br>Date | AE<br>Description | Severity<br>of AE | Related-<br>ness to<br>Oral<br>Study<br>Drug | Related-<br>ness to<br>Injectable<br>Study<br>Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| SC BHSPC | | | | | | | | | | | | |
| WS CODA,<br>Inc. | | | | | | | | | | | | |
| GNY SURC -<br>Columbia | | | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | | | |
| WS SURU -<br>SFDPH | | | | | | | | | | | | |
| TX UCLA<br>CBAM | | | | | | | | | | | | |
| TX UT Health<br>CNRA | | | | | | | | | | | | |
| TX UTSW | | | | | | | | | | | | |

## Listing 2: Non-Treatment Emergent Adverse Events in Randomized Participants by Treatment Arm Treatment Arm = Placebo/Placebo

| | | | | | | | | | | | | MedDR | A v22.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Participant ID | Random-<br>ization<br>Date | Re-ran-<br>domi-<br>zation<br>Date | Onset<br>Date | AE<br>Description | Severity of AE | Related-<br>ness to<br>Oral<br>Study<br>Drug | Related-<br>ness to<br>Injectable<br>Study<br>Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associ-<br>ated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| SC BHSPC | | | | | | | | | | | | | |
| WS CODA,<br>Inc. | | | | | | | | | | | | | |
| GNY SURC -<br>Columbia | | | | | | | | | | | | | |
| NS<br>Hennepin<br>Healthcare | | | | | | | | | | | | | |
| WS SURU -<br>SFDPH | | | | | | | | | | | | | |
| TX UCLA<br>CBAM | | | | | | | | | | | | | |
| TX UT<br>Health<br>CNRA | | | | | | | | | | | | | |
| TX UTSW | | | | | | | | | | | | | |

## Listing 2: Non-Treatment Emergent Adverse Events in Randomized Participants by Treatment Arm Treatment Arm = Placebo/AMC

| | | | | | | | | | | | | MedDR | A v22.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Participant ID | Random-<br>ization<br>Date | Re-ran-<br>domi-<br>zation-<br>Date | Onset<br>Date | AE<br>Description | Severity of AE | Related-<br>ness to<br>Oral<br>Study<br>Drug | Related-<br>ness to<br>Injectable<br>Study<br>Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associ-<br>ated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| SC BHSPC | | | | | | | | | | | | | |
| WS CODA,<br>Inc. | | | | | | | | | | | | | |
| GNY SURC -<br>Columbia | | | | | | | | | | | | | |
| NS<br>Hennepin<br>Healthcare | | | | | | | | | | | | | |
| WS SURU -<br>SFDPH | | | | | | | | | | | | | |
| TX UCLA<br>CBAM | | | | | | | | | | | | | |
| TX UT<br>Health<br>CNRA | | | | | | | | | | | | | |
| TX UTSW | | | | | | | | | | | | | |

## Listing 2: Non-Treatment Emergent Adverse Events in Randomized Participants by Treatment Arm Treatment Arm = AMC

| | | | | | | | | | | | MedDR | A v22.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Participant ID | Random-<br>ization<br>Date | Onset<br>Date | AE<br>Description | Severity<br>of AE | Related-<br>ness to<br>Oral Study<br>Drug | Related-<br>ness to<br>Injectable<br>Study<br>Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| SC BHSPC | | | | | | | | | | | | |
| WS CODA,<br>Inc. | | | | | | | | | | | | |
| GNY SURC -<br>Columbia | | | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | | | |
| WS SURU -<br>SFDPH | | | | | | | | | | | | |
| TX UCLA<br>CBAM | | | | | | | | | | | | |
| TX UT Health<br>CNRA | | | | | | | | | | | | |
| TX UTSW | | | | | | | | | | | | |

| | | | | | | | | | | MedDR | A v22.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Participant ID | Onset<br>Date | AE<br>Description | Severity<br>of AE | Related-<br>ness to<br>Oral<br>Study<br>Drug | Related-<br>ness to<br>Injectable<br>Study<br>Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| SC BHSPC | | | | | | | | | | | |
| WS CODA,<br>Inc. | | | | | | | | | | | |
| GNY SURC -<br>Columbia | | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | | |
| WS SURU -<br>SFDPH | | | | | | | | | | | |
| TX UCLA<br>CBAM | | | | | | | | | | | |
| TX UT Health<br>CNRA | | | | | | | | | | | |
| TX UTSW | | | | | | | | | | | <br> |

| Table 47: Summary of Treatment Emergent Serious A by Treatment Arm in Stage 1 | dverse E | vents | |
|---|---|---|---|
| | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Number of participants with treatment emergent serious adverse events in Stage 1 <sup>1</sup> | N (%) | | |
| Number of treatment emergent serious adverse events | N | | |
| Type of treatment emergent serious adverse event | | | |
| Death | N (%) | | |
| Life-threatening event | | | |
| Inpatient admission to hospital or prolongation of existing hospitalization | | | |
| Persistent or significant incapacity | | | |
| Congenital anomaly or birth defect | | | |
| Important medical event that required intervention to prevent any of the above | | | |
| Seizure | | | |
| Relationship of treatment emergent serious adverse event to oral study medication | | | |
| No | N (%) | | |
| Yes | | | |
| Relationship of treatment emergent serious adverse event to injectable study medication | | | |
| No | N (%) | | |
| Yes | | | |

<sup>&</sup>lt;sup>1</sup> Stage 1 SAEs include serious adverse events occurring before the date of re-randomization for re-randomized participants and in Weeks 1-6 for non-re-randomized participants.

Table 48: Summary of Treatment Emergent Serious Adverse Events by Treatment Arm in Stage 2

| | Re-ran | domized | Not Re-rar | | |
|---|---|---|---|---|---|
| | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Number of participants with treatment emergent serious adverse events in Stage 2 <sup>1</sup> | N (%) | | | | |
| Number of treatment emergent serious adverse events | N | | | | |
| Type of treatment emergent serious adverse event | | | | | |
| Death | N (%) | | | | |
| Life-threatening event | | | | | |
| Inpatient admission to hospital or prolongation of existing hospitalization | | | | | |
| Persistent or significant incapacity | | | | | |
| Congenital anomaly or birth defect | | | | | |
| Important medical event that required intervention to prevent any of the above | | | | | |
| Seizure | | | | | |
| Relationship of treatment emergent serious adverse event to oral study medication | | | | | |
| No | N (%) | | | | |
| Yes | | | | | |
| Relationship of treatment emergent serious adverse event to injectable study medication | | | | | |
| No | N (%) | | | | |
| Yes | | | | | |

<sup>&</sup>lt;sup>1</sup> Stage 2 SAEs include serious adverse events occurring on or after the date of re-randomization for re-randomized participants and in Weeks 7 or greater for non-re-randomized participants.

Dehydration

| by Treatment Arr | n in Stage T | | |
|---|---|---|---|
| System Organ Class/<br>Preferred Term (MedDRA v22.0) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Psychiatric disorders | N (%) | | |
| Suicidal ideation | N (%) | | |
| Suicide attempt | | | |
| Self-injurious behavior | | | |
| Psychotic disorder | | | |
| Depression suicidal | | | |
| Depression | | | |
| Delirium | | | |
| Anxiety | | | |
| Affective disorder | | | |
| Injury, poisoning and procedural complications | N (%) | | |
| Overdose | N (%) | | |
| Multiple fractures | | | |
| Burns third degree | | | |
| Infections and infestations | N (%) | | |
| Cellulitis | N (%) | | |
| Abscess limb | | | |
| Pneumonia | | | |
| Influenza | | | |
| Groin abscess | | | |
| Gastroenteritis | | | |
| Bronchitis | | | |
| Nervous system disorders | N (%) | | |
| Syncope | N (%) | | |
| Seizure | | | |
| Facial paresis | | | |
| Respiratory, thoracic and mediastinal disorders | N (%) | | |
| Respiratory depression | N (%) | | |
| Asthma | | | |
| Musculoskeletal and connective tissue disorders | N (%) | | |
| Back pain | N (%) | | |
| Metabolism and nutrition disorders | N (%) | | |

<sup>&</sup>lt;sup>1</sup> Stage 1 SAEs include serious adverse events occurring before the date of re-randomization for re-randomized participants and in Weeks 1-6 for non-re-randomized participants.

N (%)

Table 50: Summary of Treatment Emergent MedDRA Coded Serious Adverse Events by Treatment Arm in Stage 2

| System Organ Class/<br>Preferred Term (MedDRA v22.0) | Re-randomized | | Not Re-randomized | | |
|---|---|---|---|---|---|
| | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Participants with at least one serious adverse event in Stage 2 <sup>1</sup> | N (%) | | | | |
| Psychiatric disorders | N (%) | | | | |
| Suicidal ideation | N (%) | | | | |
| Suicide attempt | | | | | |
| Self-injurious behavior | | | | | |
| Psychotic disorder | | | | | |
| Depression suicidal | | | | | |
| Depression | | | | | |
| Delirium | | | | | |
| Anxiety | | | | | |
| Affective disorder | | | | | |
| Injury, poisoning and procedural complications | N (%) | | | | |
| Overdose | N (%) | | | | |
| Multiple fractures | | | | | |
| Burns third degree | | | | | |
| Infections and infestations | N (%) | | | | |
| Cellulitis | N (%) | | | | |
| Abscess limb | | | | | |
| Pneumonia | | | | | |
| Influenza | | | | | |
| Groin abscess | | | | | |
| Gastroenteritis | | | | | |
| Bronchitis | | | | | |
| Nervous system disorders | N (%) | | | | |
| Syncope | N (%) | | | | |
| Seizure | | | | | |
| Facial paresis | | | | | |
| Respiratory, thoracic and mediastinal disorders | N (%) | | | | |
| Respiratory depression | N (%) | | | | |
| Asthma | | | | | |
| Musculoskeletal and connective tissue disorders | N (%) | | | | |
| Back pain | N (%) | | | | |

<sup>&</sup>lt;sup>1</sup> Stage 2 AEs include adverse events occurring on or after the date of re-randomization for re-randomized participants and in Weeks 7 or greater for non-re-randomized participants.
| | | | Listing 4 | | Adverse Event Arm = Not | - | | n | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | MedDR | A v22.0 |
| Treatment<br>Emergent | Participant ID | Onset<br>Date | AE<br>Description | Severity<br>of AE | Related-<br>ness to Oral<br>Study Drug | Related-<br>ness to<br>Injectable<br>Study Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| No | | | | | | | | | | | |

| | Listing 4: Serious Adverse Events by Treatment Arm Treatment Arm = Placebo | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | MedDR | A v22.0 |
| Treatment<br>Emergent | Participant ID | Random-<br>ization<br>Date | Onset<br>Date | AE<br>Description | Severity<br>of AE | Related-<br>ness to Oral<br>Study Drug | Related-<br>ness to<br>Injectable<br>Study Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| No | | | | | | | | | | | | |
| Yes | | | | | | | | | | | | |

| Listing 4: Serious Adverse Events by Treatment Arm |
|----------------------------------------------------|
| Treatment Arm = Placebo/Placebo |

| | | | | | | | | | | | | MedDRA | A v22.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Emergent | Participant ID | Random-<br>ization<br>Date | Re-<br>random-<br>ization<br>Date | Onset<br>Date | AE<br>Description | Severity<br>of AE | Related-<br>ness to Oral<br>Study Drug | Related-<br>ness to<br>Injectable<br>Study Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| No | | | | | | | | | | | | | |
| Yes | | | | | | | | | | | | | |

# Listing 4: Serious Adverse Events by Treatment Arm Treatment Arm = Placebo/AMC

| | | | | | | | | | | | | MedDR | A v22.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Emergent | Participant ID | Random-<br>ization<br>Date | ization | Onset Date | AE<br>Description | Severity<br>of AE | Related-<br>ness to Oral<br>Study Drug | Related-<br>ness to<br>Injectable<br>Study Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| No | | | | | | | | | | | | | |
| Yes | | | | | | | | | | | | | |

NIDA CTN-0068: ADAPT-2

Statistical Analysis Plan

Version 3.0

September 13, 2019

# Listing 4: Serious Adverse Events by Treatment Arm Treatment Arm = AMC

| | | | | | | | | | | | | MedDR | A v22.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Emergent | Participant ID | Random-<br>ization<br>Date | Re-<br>random-<br>ization<br>Date | Onset<br>date | AE<br>Description | Severity<br>of AE | Related-<br>ness to<br>Oral Study<br>Drug | Related-<br>ness to<br>Injectable<br>Study Drug | Outcome | Resolu-<br>tion<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ<br>Class |
| No | | | | | | | | | | | | | |
| Yes | | | | | | | | | | | | | |

| Table 51: Summary of Injection Site Abnormali | ities by Tre | eatment | Arm in |
|---|---|---|---|
| | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Number of participants with an injection site abnormality in Stage 1 <sup>1</sup> | | | |
| Number of injection site abnormalities reported | | | |
| Type of injection site abnormality | | | |
| Pain | | | |
| Tenderness | | | |
| Bruising | | | |
| Induration | | | |
| Erythema (redness) | | | |
| Hematoma | | | |
| Swelling | | | |
| Pruritus | | | |
| Other | | | |
| Cellulitis | | | |
| Warmth | | | |
| Nodule | | | |
| Abscess | | | |
| Sterile abscess | | | |
| Necrosis | | | |
| Severity of injection site abnormality | | | |
| Mild | | | |
| Moderate | | | |
| Severe | | | |

<sup>&</sup>lt;sup>1</sup>Abnormalities occurring after injection #1 and injection #2 are reported in Stage 1.

| | Re-rand | domized | Not randor | | |
|---|---|---|---|---|---|
| | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Number of participants with an injection site abnormality in Stage 2 <sup>1</sup> | N (%) | | | | |
| Number of injection site abnormalities reported | N | | | | |
| Type of injection site abnormality | | | | | |
| Pain | N (%) | | | | |
| Tenderness | | | | | |
| Bruising | | | | | |
| Induration | | | | | |
| Erythema (redness) | | | | | |
| Hematoma | | | | | |
| Swelling | | | | | |
| Pruritus | | | | | |
| Other | | | | | |
| Cellulitis | | | | | |
| Warmth | | | | | |
| Nodule | | | | | |
| Abscess | | | | | |
| Sterile abscess | | | | | |
| Necrosis | | | | | |
| Severity of injection site abnormality | | | | | |
| Mild | N (%) | | | | |
| Moderate | | | | | |
| Severe | | | | | |

<sup>&</sup>lt;sup>1</sup> Abnormalities occurring after injection #3 and injection #4 are reported in Stage 2.

# Listing 5: Injection Site Abnormalities by Treatment Arm Treatment Arm = Placebo Event Event Resolution Abnormal

| Site | Participant ID | Randomization<br>Date | Date of Injection | Injection<br>Number | Event<br>Start<br>Date | Event<br>Resolution<br>Date | Abnormal<br>Event | Severity | Treatment |
|---|---|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | | | |
| WS CODA, Inc. | | | | | | | | | |
| GNY SURC –<br>Columbia | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | |
| WS SURU – SFDPH | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | |
| TX UTSW | | | | | | | | | |

NIDA CTN-0068: ADAPT-2 Statistical Analysis Plan

# Listing 5: Injection Site Abnormalities by Treatment Arm Treatment Arm = Placebo/Placebo

| Site | Participant ID | Randomization<br>Date | Re-<br>randomization<br>Date | Date of Injection | Injection<br>Number | Event<br>Start<br>Date | Event<br>Resolution<br>Date | Abnormal<br>Event | Severity | Treatment |
|---|---|---|---|---|---|---|---|---|---|---|
| SC BHSPC | 1 | | | - | | | | | | |
| WS CODA, Inc. | | | | | | | | | | |
| GNY SURC –<br>Columbia | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | |
| WS SURU – SFDPH | | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | | |
| TX UTSW | | | | | | | | | | |

NIDA CTN-0068: ADAPT-2 Statistical Analysis Plan

# Listing 5: Injection Site Abnormalities by Treatment Arm Treatment Arm = Placebo/AMC

| Site | Participant ID | Randomization<br>Date | Re-<br>randomization<br>Date | Date of Injection | Injection<br>Number | Event<br>Start<br>Date | Event<br>Resolution<br>Date | Abnormal<br>Event | Severity | Treatment |
|---|---|---|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | | | | |
| WS CODA, Inc. | | | | | | | | | | |
| GNY SURC –<br>Columbia | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | |
| WS SURU – SFDPH | | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | | |
| TX UTSW | | | | | | | | | | |

# Listing 5: Injection Site Abnormalities by Treatment Arm Treatment Arm = AMC

| Site | Participant ID | Randomization<br>Date | Date of<br>Injection | Injection<br>Number | Event<br>Start<br>Date | Event<br>Resolution<br>Date | Abnormal<br>Event | Severity | Treatment |
|---|---|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | | | |
| WS CODA, Inc. | | | | | | | | | |
| GNY SURC –<br>Columbia | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | |
| WS SURU –<br>SFDPH | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | |
| TX UT Health<br>CNRA | | | | | | | | | |
| TX UTSW | | | | | | | | | |

# Listing 6: Elevated LFTs by Treatment Arm Treatment Arm = Placebo

| Site | Participant ID | Randomization<br>Date | Date of<br>Lab<br>Collection | Visit | Aspartate<br>Aminotransferase<br>(IU/L) | Alanine<br>Aminotransferase<br>(IU/L) | Total<br>Bilirubin<br>(mg/dL) |
|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | |
| WS CODA, Inc. | | | | | | | |
| GNY SURC - Columbia | | | | | | | |
| NS Hennepin Healthcare | | | | | | | |
| WS SURU - SFDPH | | | | | | | |
| TX UCLA CBAM | | | | | | | |
| TX UT Health CNRA | | | | | | | |
| TX UTSW | | | | | | | |

Lab values above thresholds are highlighted in yellow. This includes ALT values higher than 250 IU/L based on 5x ULN, AST values higher than 250 IU/L based on 5x ULN, and total bilirubin values higher than 2.2 mg/dL based on 2x ULN.

# Listing 6: Elevated LFTs by Treatment Arm Treatment Arm = Placebo/Placebo

| Site | Participant ID | Randomization<br>Date | Re-<br>randomization<br>Date | Date of<br>Lab<br>Collection | Visit | Aspartate<br>Aminotransferase<br>(IU/L) | Alanine<br>Aminotransferase<br>(IU/L) | Total<br>Bilirubin<br>(mg/dL) |
|---|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | | |
| WS CODA, Inc. | | | | | | | | |
| GNY SURC - Columbia | | | | | | | | |
| NS Hennepin Healthcare | | | | | | | | |
| WS SURU - SFDPH | | | | | | | | |
| TX UCLA CBAM | | | | | | | | |
| TX UT Health CNRA | | | | | | | | |
| TX UTSW | | | | | | | | |

Lab values above thresholds are highlighted in yellow. This includes ALT values higher than 250 IU/L based on 5x ULN, AST values higher than 250 IU/L based on 5x ULN, and total bilirubin values higher than 2.2 mg/dL based on 2x ULN.

# Listing 6: Elevated LFTs by Treatment Arm Treatment Arm = Placebo/AMC

| Site | Participant ID | Randomization<br>Date | Re-<br>randomization<br>Date | Date of<br>Lab<br>Collection | Visit | Aspartate<br>Aminotransferase<br>(IU/L) | Alanine<br>Aminotransferase<br>(IU/L) | Total<br>Bilirubin<br>(mg/dL) |
|---|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | | |
| WS CODA, Inc. | | | | | | | | |
| GNY SURC - Columbia | | | | | | | | |
| NS Hennepin Healthcare | | | | | | | | |
| WS SURU - SFDPH | | | | | | | | |
| TX UCLA CBAM | | | | | | | | |
| TX UT Health CNRA | | | | | | | | |
| TX UTSW | | | | | | | | |

Lab values above thresholds are highlighted in yellow. This includes ALT values higher than 250 IU/L based on 5x ULN, AST values higher than 250 IU/L based on 5x ULN, and total bilirubin values higher than 2.2 mg/dL based on 2x ULN.

# Listing 6: Elevated LFTs by Treatment Arm Treatment Arm = AMC

| Site | Participant ID | Randomization<br>Date | Date of<br>Lab<br>Collection | Visit | Aspartate<br>Aminotransferase<br>(IU/L) | Alanine<br>Aminotransferase<br>(IU/L) | Total<br>Bilirubin<br>(mg/dL) |
|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | (1012) | (1012) | (3) |
| WS CODA, Inc. | | | | | | | |
| GNY SURC - Columbia | | | | | | | |
| NS Hennepin Healthcare | | | | | | | |
| WS SURU - SFDPH | | | | | | | |
| TX UCLA CBAM | | | | | | | |
| TX UT Health CNRA | | | | | | | |
| TX UTSW | | | | | | | |

Lab values above thresholds are highlighted in yellow. This includes ALT values higher than 250 IU/L based on 5x ULN, AST values higher than 250 IU/L based on 5x ULN, and total bilirubin values higher than 2.2 mg/dL based on 2x ULN.

| Listing 7: Decreased Platelets by Treatment Arm Treatment Arm = Placebo | |
|---|---|
| Site | Participant ID Date of Collection Visit Platelets (μ |
| SC BHSPC | |
| WS CODA, Inc. | |
| GNY SURC - Columbia | |
| NS Hennepin Healthcare | |
| WS SURU - SFDPH | |
| TX UCLA CBAM | |
| TX UT Health CNRA | |
| TX UTSW | |

Platelet values under the threshold of 75x10<sup>3</sup>/µL are highlighted in yellow.

All visits are included for participants who experienced decreased platelets at any visit.

| Listing 7: Decreased Platelets by Treatment Arm Treatment Arm = Placebo/Placebo |
|---|
| Re-randomization Date Date of Lab Collection Visit Platelets (μL) |
| SC BHSPC |
| WS CODA, Inc. |
| GNY SURC - Columbia |
| NS Hennepin Healthcare |
| WS SURU - SFDPH |
| TX UCLA CBAM |
| TX UT Health CNRA |
| TX UTSW |

Platelet values under the threshold of 75x10<sup>3</sup>/µL are highlighted in yellow.

All visits are included for participants who experienced decreased platelets at any visit.

| Listing 7: Decreased Platelets by Treatment Arm Treatment Arm = Placebo/AMC |
|---|
| Randomization Date Participant ID Participant ID Date Participant ID Date Platelets (μL) |
| SC BHSPC |
| WS CODA, Inc. |
| GNY SURC - Columbia |
| NS Hennepin Healthcare |
| WS SURU - SFDPH |
| TX UCLA CBAM |
| TX UT Health CNRA |
| TX UTSW |

Platelet values under the threshold of 75x10<sup>3</sup>/µL are highlighted in yellow.

All visits are included for participants who experienced decreased platelets at any visit.

| Listing 7: Decreased Platelets by Treatment Arm Treatment Arm = AMC |
|---|
| Site Participant ID Randomization Date Of Lab Collection Visit Platelets (μ |
| SC BHSPC |
| WS CODA, Inc. |
| GNY SURC - Columbia |
| NS Hennepin Healthcare |
| WS SURU - SFDPH |
| TX UCLA CBAM |
| TX UT Health CNRA |
| TX UTSW |

Platelet values under the threshold of 75x10<sup>3</sup>/µL are highlighted in yellow.

All visits are included for participants who experienced decreased platelets at any visit.

| Table 53: Summary of Elevated QTc Intervals by Treatment Arm | | | | | |
|---|---|---|---|---|---|
| | Re-randomized | | Not Re-rai | ndomized | |
| | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Participants with elevated QTc intervals ≥ 500 ms at Week 12 | n/N (%) | | | | |
| Baseline QTc interval (ms) | | | | | |
| N | | | | | |
| Mean | | | | | |
| SD | | | | | |
| Min | | | | | |
| 25th percentile | | | | | |
| Median | | | | | |
| 75th percentile | | | | | |
| Max | | | | | |
| Week 12 QTc interval (ms) | | | | | |
| N | | | | | |
| Mean | | | | | |
| SD | | | | | |
| Min | | | | | |
| 25th percentile | | | | | |
| Median | | | | | |
| 75th percentile | | | | | |
| Max | | | | | |

| | Re-rand | lomized | Not Re-rar | ndomized | |
|---|---|---|---|---|---|
| | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) | Total<br>(N=) |
| Change from baseline QTc interval (ms) at Week 12 | | | | | |
| N | | | | | |
| Mean | | | | | |
| SD | | | | | |
| Min | | | | | |
| 25th percentile | | | | | |
| Median | | | | | |
| 75th percentile | | | | | |
| Max | | | | | |

| Listing 8: AV Block ECG Abnormalities by Treatment Arm Treatment Arm = Placebo |
|---|
| Randomization Date of ECG Week 12 Second Degree AV Block Present Present Present |
| SC BHSPC |
| WS CODA, Inc. |
| GNY SURC - Columbia |
| NS Hennepin Healthcare |
| WS SURU - SFDPH |
| TX UCLA CBAM |
| TX UT Health CNRA |
| TX UTSW |

| Listing 8: AV Block ECG Abnormalities by Treatment Arm Treatment Arm = Placebo/Placebo |
|---|
| Randomization Date Re-randomi- zation Date Re- randomi- zation Date Re- randomi- zation Date Re- randomi- zation Date Re- randomi- zation Date Re- randomi- zation Date Date of ECG Week 12 Second Degree AV Block Present Present |
| SC BHSPC |
| WS CODA, Inc. |
| GNY SURC - Columbia |
| NS Hennepin Healthcare |
| WS SURU - SFDPH |
| TX UCLA CBAM |
| TX UT Health CNRA |
| TX UTSW |

TX UT Health CNRA

TX UTSW

# Listing 8: AV Block ECG Abnormalities by Treatment Arm Treatment Arm = Placebo/AMC

| Site | Participant ID | Randomization<br>Date | Re-<br>randomi-<br>zation Date | Date of ECG | Week 12 Second<br>Degree AV Block<br>Present | Week 12 Third<br>Degree AV Block<br>Present |
|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | |
| WS CODA, Inc. | | | | | | |
| GNY SURC - Columbia | | | | | | |
| NS Hennepin Healthcare | | | | | | |
| WS SURU - SFDPH | | | | | | |
| TX UCLA CBAM | | | | | | |
| TX UT Health CNRA | | | | | | |
| TX UTSW | | | | | | |

| Listing | Listing 8: AV Block ECG Abnormalities by Treatment Arm Treatment Arm = AMC | | | | |
|---|---|---|---|---|---|
| Site | Participant ID | Randomization<br>Date | Date of<br>ECG | Week 12<br>Second<br>Degree AV<br>Block<br>Present | Week 12 Third<br>Degree AV<br>Block Present |
| SC BHSPC | | | | | |
| WS CODA, Inc. | | | | | |
| GNY SURC - Columbia | | | | | |
| NS Hennepin Healthcare | | | | | |
| WS SURU - SFDPH | | | | | |
| TX UCLA CBAM | | | | | |

| Table 54: Summary of Suicide Risk by Treatment Arm in Stage 1 | | |
|---|---|---|
| | AMC<br>(N=) | Total<br>(N=) |
| Number endorsing on CHRT or PHQ-9 | N (%) | |
| Number endorsing on CHRT only | N (%) | |
| Number endorsing on PHQ-9 only | N (%) | |
| Number endorsing on CHRT and PHQ-9 | N (%) | |

Endorsing suicide risk on CHRT is defined as responses of Agree or Strongly Agree on any of CHRT questions 13, 14, or 15. Endorsing suicide risk on PHQ-9 is defined as responses of Several Days or More than Half the Days or Nearly Every Day to PHQ-9 question 9.

| Table 55: Summary of Suicide Risk by Treatment Arm in Stage 2 | | | | |
|---|---|---|---|---|
| | Re-randomized Not Re-randomize | | | |
| | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) |
| Number endorsing on CHRT or PHQ-9 | N (%) | | | |
| Number endorsing on CHRT only | N (%) | | | |
| Number endorsing on PHQ-9 only | N (%) | | | |
| Number endorsing on CHRT and PHQ-9 | N (%) | | | |

Endorsing suicide risk on CHRT is defined as responses of Agree or Strongly Agree on any of CHRT questions 13, 14, or 15. Endorsing suicide risk on PHQ-9 is defined as responses of Several Days or More than Half the Days or Nearly Every Day to PHQ-9 question 9.

| Table 56: Summary of Suicide Risk by Treatment Arm in Follow-up Period | | | | |
|---|---|---|---|---|
| | Re-randomized Not Re-randomized | | | |
| | Placebo/<br>Placebo<br>(N=) | Placebo/<br>AMC<br>(N=) | Placebo<br>(N=) | AMC<br>(N=) |
| Number endorsing on CHRT or PHQ-9 | N (%) | | | |
| Number endorsing on CHRT only | N (%) | | | |
| Number endorsing on PHQ-9 only | N (%) | | | |
| Number endorsing on CHRT and PHQ-9 | N (%) | | | |

Endorsing suicide risk on CHRT is defined as responses of Agree or Strongly Agree on any of CHRT questions 13, 14, or 15. Endorsing suicide risk on PHQ-9 is defined as responses of Several Days or More than Half the Days or Nearly Every Day to PHQ-9 question 9.

TX UTSW

#### **Listing 9: Suicide Risk by Treatment Arm Treatment Arm = Placebo CHRT** PHQ-9 I Have Thoughts about Thoughts You are I Have Been Having Thoughts of Killing How I Might Kill I Have a Plan to Kill Better Off Dead or **Participant ID** Myself Myself of Hurting Yourself Site Visit Myself SC BHSPC WS CODA, Inc. GNY SURC - Columbia NS Hennepin Healthcare WS SURU - SFDPH TX UCLA CBAM TX UT Health CNRA

All visits are included for participants who endorsed suicide risk at any visit on either CHRT or PHQ-9.

### **Listing 9: Suicide Risk by Treatment Arm Treatment Arm = Placebo/Placebo CHRT** PHQ-9 I Have Thoughts about Thoughts You are I Have Been Having Thoughts of Killing How I Might Kill I Have a Plan to Kill Better Off Dead or **Participant ID** Myself of Hurting Yourself Site Visit Myself Myself SC BHSPC WS CODA, Inc. GNY SURC - Columbia NS Hennepin Healthcare WS SURU - SFDPH TX UCLA CBAM TX UT Health CNRA TX UTSW

All visits are included for participants who were endorse suicide risk at any visit on either CHRT or PHQ-9.

### Listing 9: Suicide Risk by Treatment Arm **Treatment Arm = Placebo/AMC CHRT** PHQ-9 I Have Thoughts about Thoughts You are I Have Been Having Thoughts of Killing How I Might Kill I Have a Plan to Kill Better Off Dead or **Participant ID** Myself Myself of Hurting Yourself Site Visit Myself SC BHSPC WS CODA, Inc. GNY SURC - Columbia NS Hennepin Healthcare WS SURU - SFDPH TX UCLA CBAM TX UT Health CNRA TX UTSW

All visits are included for participants who were endorse suicide risk at any visit on either CHRT or PHQ-9.

| Listing 9: Suicide Risk by Treatment Arm Treatment Arm = AMC | | | | | | |
|---|---|---|---|---|---|---|
| | | | | CHRT | | PHQ-9 |
| Site | Participant ID | Visit | l Have Been Having<br>Thoughts of Killing<br>Myself | I Have Thoughts about<br>How I Might Kill<br>Myself | l Have a Plan to Kill<br>Myself | Thoughts You are<br>Better Off Dead or<br>of Hurting Yourself |
| SC BHSPC | | | | | | |
| WS CODA, Inc. | | | | | | |
| GNY SURC - Columbia | | | | | | |
| NS Hennepin Healthcare | | | | | | |
| WS SURU - SFDPH | | | | | | |
| TX UCLA CBAM | | | | | | |
| TX UT Health CNRA | | | | | | |
| TX UTSW | | | | | | |

All visits are included for participants who were endorse suicide risk at any visit on either CHRT or PHQ-9.

# Listing 10: Pregnancies by Treatment Arm Treatment Arm = Placebo

| | Doublein out | Date of | Date Staff | Date | Date of Last<br>Dose of Oral | Date of Last | Danasanasa | Date of | Normal |
|---|---|---|---|---|---|---|---|---|---|
| Site | Participant<br>ID | Randomization | Aware of<br>Pregnancy | Pregnancy<br>Confirmed | Study<br>Medication | Injectable Study<br>Medication | Pregnancy<br>Outcome | Pregnancy<br>Outcome | Infant? |
| SC BHSPC | | | | | | | | | |
| WS CODA,<br>Inc. | | | | | | | | | |
| GNY SURC -<br>Columbia | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | |
| WS SURU -<br>SFDPH | | | | | | | | | |
| TX UCLA<br>CBAM | | | | | | | | | |
| TX UT Health<br>CNRA | | | | | | | | | |
| TX UTSW | | | | | | | | | |

# Listing 10: Pregnancies by Treatment Arm Treatment Arm = Placebo/Placebo

| | ı | I | I I | | I | | 1 | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Site | Participant<br>ID | Date of<br>Randomization | Date of Re-<br>randomization | Date Staff<br>Aware of<br>Pregnancy | Date<br>Pregnancy<br>Confirmed | Date of Last<br>Dose of Oral<br>Study<br>Medication | Date of Last<br>Injectable Study<br>Medication | Pregnancy<br>Outcome | Date of<br>Pregnancy<br>Outcome | Normal<br>Infant? |
| SC BHSPC | | | | | | | | | | |
| WS CODA,<br>Inc. | | | | | | | | | | |
| GNY SURC -<br>Columbia | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | |
| WS SURU -<br>SFDPH | | | | | | | | | | |
| TX UCLA<br>CBAM | | | | | | | | | | |
| TX UT Health<br>CNRA | | | | | | | | | | |
| TX UTSW | | | | | | | | | | |

# Listing 10: Pregnancies by Treatment Arm Treatment Arm = Placebo/AMC

| | ı | I | I I | | I | | 1 | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Site | Participant<br>ID | Date of<br>Randomization | Date of Re-<br>randomization | Date Staff<br>Aware of<br>Pregnancy | Date<br>Pregnancy<br>Confirmed | Date of Last<br>Dose of Oral<br>Study<br>Medication | Date of Last<br>Injectable Study<br>Medication | Pregnancy<br>Outcome | Date of<br>Pregnancy<br>Outcome | Normal<br>Infant? |
| SC BHSPC | | | | | | | | | | |
| WS CODA,<br>Inc. | | | | | | | | | | |
| GNY SURC -<br>Columbia | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | |
| WS SURU -<br>SFDPH | | | | | | | | | | |
| TX UCLA<br>CBAM | | | | | | | | | | |
| TX UT Health<br>CNRA | | | | | | | | | | |
| TX UTSW | | | | | | | | | | |

# Listing 10: Pregnancies by Treatment Arm Treatment Arm = AMC

| Site | Participant<br>ID | Date of<br>Randomization | Date Staff<br>Aware of<br>Pregnancy | Date<br>Pregnancy<br>Confirmed | Date of Last<br>Dose of Oral<br>Study<br>Medication | Date of Last<br>Injectable Study<br>Medication | Pregnancy<br>Outcome | Date of<br>Pregnancy<br>Outcome | Normal<br>Infant? |
|---|---|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | | | |
| WS CODA,<br>Inc. | | | | | | | | | |
| GNY SURC -<br>Columbia | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | |
| WS SURU -<br>SFDPH | | | | | | | | | |
| TX UCLA<br>CBAM | | | | | | | | | |
| TX UT Health<br>CNRA | | | | | | | | | |
| TX UTSW | | | | | | | | | |

### **Listing 11: Deaths by Treatment Arm Treatment Arm = Placebo** MedDRA v22.0 Randomization Preferred System Organ Class Site Participant ID Description Date **Date of Death** Term SC BHSPC WS CODA, Inc. GNY SURC - Columbia NS Hennepin Healthcare WS SURU - SFDPH TX UCLA CBAM TX UT Health CNRA TX UTSW

# Listing 11: Deaths by Treatment Arm Treatment Arm = Placebo/Placebo

| Site | | | Re- | | | MedDF | RA v22.0 |
|---|---|---|---|---|---|---|---|
| | Participant ID | Randomization<br>Date | randomization<br>Date | Date of Death | Description | Preferred<br>Term | System<br>Organ Class |
| SC BHSPC | | | | | | | |
| WS CODA, Inc. | | | | | | | |
| GNY SURC - Columbia | | | | | | | |
| NS Hennepin Healthcare | | | | | | | |
| WS SURU - SFDPH | | | | | | | |
| TX UCLA CBAM | | | | | | | |
| TX UT Health CNRA | | | | | | | |
| TX UTSW | | | | | | | |

# Listing 11: Deaths by Treatment Arm Treatment Arm = Placebo/AMC

| Site | | | Do. | | | MedDF | MedDRA v22.0 |
|---|---|---|---|---|---|---|---|
| | Participant ID | Randomization<br>Date | Re-<br>randomization<br>Date | Date of Death | Description | Preferred<br>Term | System<br>Organ Class |
| SC BHSPC | | | | | | | |
| WS CODA, Inc. | | | | | | | |
| GNY SURC - Columbia | | | | | | | |
| NS Hennepin Healthcare | | | | | | | |
| WS SURU - SFDPH | | | | | | | |
| TX UCLA CBAM | | | | | | | |
| TX UT Health CNRA | | | | | | | |
| TX UTSW | | | | | | | |

TX UTSW

### **Listing 11: Deaths by Treatment Arm Treatment Arm = AMC** MedDRA v22.0 Randomization Preferred System **Date of Death** Organ Class Site Participant ID Description Date Term SC BHSPC WS CODA, Inc. GNY SURC - Columbia NS Hennepin Healthcare WS SURU - SFDPH TX UCLA CBAM TX UT Health CNRA

| | Table 57 | : Summary of | Data Audits | |
|---|---|---|---|---|
| Site | Date of<br>Audit | Total Fields<br>Audited <sup>1</sup> | Total Data<br>Discrepancies <sup>2</sup> | Error Rate (%) |
| SC BHSPC | | | | |
| | Subtotal | | | |
| WS CODA, Inc. | | | | |
| | Subtotal | | | |
| GNY SURC - Columbia | | | | |
| | Subtotal | | | |
| NS Hennepin Healthcare | | | | |
| | Subtotal | | | |
| WS SURU - SFDPH | | | | |
| | Subtotal | | | |
| TX UCLA CBAM | | | | |
| | Subtotal | | | |
| TX UT Health CNRA | | | | |
| | Subtotal | | | |
| TX UTSW | | | | |
| | Subtotal | | | |
| Total | | | | |

<sup>&</sup>lt;sup>1</sup> Fields reviewed at monitoring visit comparing the database to source documentation.

<sup>&</sup>lt;sup>2</sup> Fields discrepant between database and source documentation.

| Ta | able 58: S | ummary o | of Protocol | Deviation | s | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | SC<br>BHSPC | WS<br>CODA,<br>Inc. | GNY<br>SURC -<br>Columbia | NS<br>Hennepin<br>Healthcare | WS SURU<br>- SFDPH | TX UCLA<br>CBAM | TX UT<br>Health<br>CNRA | TX UTSW | Total |
| Total number of protocol deviations | N | | | | | | | | |
| Number of participants impacted per protocol deviation | | | | | | | | | |
| None | N (%) | | | | | | | | |
| One | | | | | | | | | |
| More than one | | | | | | | | | |
| Total number of major protocol deviations | N | | | | | | | | |
| Type of major protocol deviation | | | | | | | | | |
| Safety assessment (e.g. labs, ECG, clinical referral to care) not conducted per protocol | N (%) | | | | | | | | |
| Medication dosing errors (protocol specified dose not dispensed) | | | | | | | | | |
| Total number of minor protocol deviations | N | | | | | | | | |
| Type of minor protocol deviation | | | | | | | | | |
| AE/SAE reported out of protocol specified reporting timeframe | N (%) | | | | | | | | |
| Biologic specimen not collected/processed as per protocol | | | | | | | | | |
| Study assessments not completed/followed as per protocol | | | | | | | | | |
| Study medication management - Other | | | | | | | | | |
| Other study procedures/assessments issues | | | | | | | | | |
| Informed consent/assent process not properly conducted and/or documented | | | | | | | | | |
| Other significant deviations issues | | | | | | | | | |
| Protocol required visit/assessment not scheduled or conducted | | | | | | | | | |
| Other informed consent/assent procedures issues | | | | | | | | | |
| AE not reported | | | | | | | | | |
| Other inclusion/exclusion criteria issues | | | | | | | | | |
| Other study devices issues | | | | | | | | | |
| Non IRB approved/outdated/obsolete informed consent/assent documents used | | | | | | | | | |
| AE/SAE not elicited, observed and/or documented as per protocol | | | | | | | | | |

# Listing 12: Listing of Protocol Deviations Deviation Category = Informed consent procedures

| Site | Related<br>Participant IDs | Date of<br>Protocol<br>Deviation | Date Protocol Deviation Entered in eClinical | Deviation<br>Type | Deviation<br>Type (other) | Deviation<br>Description | Resolution<br>Corrective<br>Action | IRB<br>Reporting<br>Required? | IRB<br>Notified<br>at<br>Continuing<br>Review? | Expected/<br>Actual<br>IRB<br>Report<br>date |
|---|---|---|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | | | | |
| WS CODA, Inc. | | | | | | | | | | |
| GNY SURC – Columbia | | | | | | | | | | |
| NS Hennepin Healthcare | | | | | | | | | | |
| WS SURU – SFDPH | | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | | |
| TX UTSW | | | | | | | | | | |

# Listing 12: Listing of Protocol Deviations Deviation Category = Inclusion/exclusion criteria

| Site | Related<br>Participant IDs | Date of<br>Protocol<br>Deviation | Date Protocol Deviation Entered in eClinical | Deviation<br>Type | Deviation<br>Type (other) | Deviation<br>Description | Resolution<br>Corrective<br>Action | IRB<br>Reporting<br>Required? | IRB Notified at Continuing Review? | Expected/<br>Actual<br>IRB<br>Report<br>date |
|---|---|---|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | | | | |
| WS CODA, Inc. | | | | | | | | | | |
| GNY SURC –<br>Columbia | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | |
| WS SURU – SFDPH | | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | | |
| TX UTSW | | | | | | | | | | |

# Listing 12: Listing of Protocol Deviations Deviation Category = Laboratory Assessments

| | | Date of | Date<br>Protocol<br>Deviation<br>Entered | | | | Resolution | IRB | IRB<br>Notified<br>at | Expected/<br>Actual<br>IRB |
|---|---|---|---|---|---|---|---|---|---|---|
| Site | Related<br>Participant IDs | Protocol<br>Deviation | in<br>eClinical | Deviation<br>Type | Deviation<br>Type (other) | Deviation<br>Description | Corrective<br>Action | Reporting Required? | Continuing Review? | Report<br>date |
| SC BHSPC | | | | | | | | | | |
| WS CODA, Inc. | | | | | | | | | | |
| GNY SURC –<br>Columbia | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | |
| WS SURU – SFDPH | | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | | |
| TX UTSW | | | | | | | | | | |

# Listing 12: Listing of Protocol Deviations Deviation Category = Study Procedures/Assessments

| | | | | | _ | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Site | Related<br>Participant IDs | Date of<br>Protocol<br>Deviation | Date Protocol Deviation Entered in eClinical | Deviation<br>Type | Deviation<br>Type (other) | Deviation<br>Description | Resolution<br>Corrective<br>Action | IRB<br>Reporting<br>Required? | IRB<br>Notified<br>at<br>Continuing<br>Review? | Expected/<br>Actual<br>IRB<br>Report<br>date |
| SC BHSPC | | | | | | | | | | |
| WS CODA, Inc. | | | | | | | | | | |
| GNY SURC –<br>Columbia | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | |
| WS SURU – SFDPH | | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | | |
| TX UTSW | | | | | | | | | | |

# Listing 12: Listing of Protocol Deviations Deviation Category = Adverse Event

| Site | Related<br>Participant IDs | Date of<br>Protocol<br>Deviation | Date<br>Protocol<br>Deviation<br>Entered<br>in<br>eClinical | Deviation<br>Type | Deviation<br>Type (other) | Deviation<br>Description | Resolution<br>Corrective<br>Action | IRB<br>Reporting<br>Required? | IRB Notified at Continuing Review? | Expected/<br>Actual<br>IRB<br>Report<br>date |
|---|---|---|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | | | | |
| WS CODA, Inc. | | | | | | | | | | |
| GNY SURC –<br>Columbia | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | |
| WS SURU – SFDPH | | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | | |
| TX UTSW | | | | | | | | | | |

# Listing 12: Listing of Protocol Deviations Deviation Category = Study Medication Management

| Site | Related<br>Participant IDs | Date of<br>Protocol<br>Deviation | Date Protocol Deviation Entered in eClinical | Deviation<br>Type | Deviation<br>Type (other) | Deviation<br>Description | Resolution<br>Corrective<br>Action | IRB<br>Reporting<br>Required? | IRB Notified at Continuing Review? | Expected/<br>Actual<br>IRB<br>Report<br>date |
|---|---|---|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | | | | |
| WS CODA, Inc. | | | | | | | | | | |
| GNY SURC –<br>Columbia | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | |
| WS SURU – SFDPH | | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | | |
| TX UTSW | | | | | | | | | | |

# Listing 12: Listing of Protocol Deviations Deviation Category = Study Devices

| Site | Related<br>Participant IDs | Date of<br>Protocol<br>Deviation | Date Protocol Deviation Entered in eClinical | Deviation<br>Type | Deviation<br>Type (other) | Deviation<br>Description | Resolution<br>Corrective<br>Action | IRB<br>Reporting<br>Required? | IRB Notified at Continuing Review? | Expected/<br>Actual<br>IRB<br>Report<br>date |
|---|---|---|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | | | | |
| WS CODA, Inc. | | | | | | | | | | |
| GNY SURC –<br>Columbia | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | |
| WS SURU – SFDPH | | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | | |
| TX UTSW | | | | | | | | | | |

# Listing 12: Listing of Protocol Deviations Deviation Category = Other Significant Deviations

| Site | Related<br>Participant IDs | Date of<br>Protocol<br>Deviation | Date Protocol Deviation Entered in eClinical | Deviation<br>Type | Deviation<br>Type (other) | Deviation<br>Description | Resolution<br>Corrective<br>Action | IRB<br>Reporting<br>Required? | IRB Notified at Continuing Review? | Expected/<br>Actual<br>IRB<br>Report<br>date |
|---|---|---|---|---|---|---|---|---|---|---|
| SC BHSPC | | | | | | | | | | |
| WS CODA, Inc. | | | | | | | | | | |
| GNY SURC –<br>Columbia | | | | | | | | | | |
| NS Hennepin<br>Healthcare | | | | | | | | | | |
| WS SURU – SFDPH | | | | | | | | | | |
| TX UCLA CBAM | | | | | | | | | | |
| TX UT Health CNRA | | | | | | | | | | |
| TX UTSW | | | | | | | | | | |